## Study Protocol and Statistical Analysis Plan

# **Proxalutamide Treatment for Hospitalized COVID-19 Patients**

| Protocol: | KP-DRUG-SARS-003 |
|--------------|-------------------------------------------------|
| Date: | 01 February, 2021 |
| EDMS number: | Brazilian National Ethics Committee (4.513.425) |
| NCT number: | NCT04728802 |

#### **Document Contents:**

#### 1. Original protocol

Note: A protocol planned for males, begins with protocol version 1.0.

- 2. Final protocol (v8) with summary of all changes.
- 3. Final statistical analysis plan with summary of all changes.

#### **Confidentiality Statement**

The information contained in this document is confidential and proprietary to the principal investigator. It is offered with the express agreement that you will not disclose this document to any other person(s), or discuss the information contained herein or make reproduction by any means electronic or mechanical, or use it for any purpose other than the evaluation of the proposed clinical study for approval by an Institutional Review Board.



# CLINICAL STUDY PROTOCOL

Proxalutamide (GT0918)
Treatment for Hospitalized
COVID-19 Male Patients

#### **Proprietary and Confidential**

The information contained in this document is confidential and proprietary to Applied Biology, Inc. It is offered with the express agreement that you will not disclose this document to any other person(s), or discuss the information contained herein or make reproduction by any means electronic or mechanical, or use it for any purpose other than the evaluation of the proposed clinical study for approval by an Institutional Review Board.



 $2 \mid P \text{ a g e}$ 

#### **PROTOCOL NAME:**

Clinical Study: Proxalutamide Treatment for Hospitalized COVID-19 Male Patients

## PROTOCOL IDENTIFYING NUMBER:

KP-DRUG-SARS-003

#### PROTOCOL VERSION NUMBER:

1.00

#### **PROTOCOL VERSION DATE:**

December 27, 2020



#### **GENERAL INFORMATION**

#### Name and address of the person(s) authorized to sign the protocol and amendments

Andy Goren, MD Flavio A. Cadegiani, MD, MSc, PhD Carlos Wambier, MD

#### Name and address of study monitor

Carlos Wambier, MD

Name, title, address and telephone number(s) of the medical expert for the trial



## Name and title of the investigator(s) and sub-investigators responsible for the trial with address and phone number(s)

Flavio A. Cadegiani, MD, MSc, PhD Andy Goren, MD Carlos Wambier, MD

#### Principal Investigator (s)

Flavio A. Cadegiani, MD, MSc, PhD Andy Goren, MD

#### **Site Supervisor**

Andy Goren, MD

#### **Investigator Assistant**

**TBD** 



4 | Page

## Protocol signature page Investigator's Agreement

Clinical Study: Proxalutamide Treatment for Hospitalized COVID-19 Male Patients

The information contained in this document is CONFIDENTIAL and, except to the extent necessary to obtain informed consent, may not be disclosed unless such disclosure is required by government regulation or state/local customs or law. Persons to whom the information is disclosed must be informed that the information is CONFIDENTIAL and not be further disclosed by them. By my signature below I agree to conduct this clinical study in accordance with the protocol, Good Clinical Practice, the Declaration of Helsinki, government regulations and state/local customs or laws, including those applying to institutional/ethics review and informed consent. I have read the protocol. I agree to ensure the confidentiality of my patients; however I agree to make available to the CROs, the Sponsor of this clinical study, relevant regulatory authorities, my patients' medical records. I am aware of my responsibilities as investigator as provided to me by the CROs.

| Name | Signature | Date |
|-----------------------------------|-----------|------|
| Flavio A. Cadegiani, MD, MSc, PhD | | |
| Andy Goren, MD | | |





## **TABLE OF CONTENTS**

| 1. | BACK | GROUND | 1 |
|----|--------|---------------------------------------------|----|
| | 1. ( | Overview | 1 |
| | 1.1. | Investigational Drug | 2 |
| | 1.1. | Pre-Clinical and Prior Clinical Data | 3 |
| | 1.1.1. | Prior Pre-Clinical and Clinical Safety Data | 3 |
| | 1.2. | Risks/Benefits | 14 |
| | 1.3. | Trial Conduct | 15 |
| | 1.4. | Population | 15 |
| | 1.5. | Literature | 15 |
| 2. | TRIAL | OBJECTIVES | 17 |
| 3. | TRIAL | DESIGN | 17 |
| | 3.1 | Primary Study Endpoints/Secondary Endpoints | 17 |
| | 3.2 | Study Design/Type | 17 |
| | 3.3 | Randomization | 18 |
| | 3.4 | Records | 19 |
| | 3.5 | Duration | 19 |
| | 3.6 | Discontinuation | 19 |
| | 3.7 | Product Accountability | 19 |
| | 3.8 | Data Identification | 20 |
| 4. | SELEC | CTION AND WITHDRAWAL OF SUBJECTS | 20 |
| | 4.1 | Inclusion Criteria | 20 |
| | 4.2 | Exclusion Criteria | 20 |



| | 4.3 | Subject Withdrawal | 6 P a g e<br>21 |
|---|---|---|---|
| | 4.4 | Treatment of Subjects | 21 |
| | 4.5 | Medication | 21 |
| 5 | 4.6<br>ASSES | Monitoring for subject compliance SSMENT OF EFFICACY | 21<br>22 |
| | 5.1 | Efficacy Parameters | 22 |
| | 5.2 | Method and Timing | 22 |
| 6 | | SSMENT OF SAFETY | |
| | 6.1 | Safety Parameters | 23 |
| | 6.2 | Method and Timing | 23 |
| | 6.3 | Adverse Event Reporting | 23 |
| | 6.4 | Definitions | 24 |
| | 6.5 | Adverse Event Follow-up | 25 |
| 7 | STAT | ISTICAL PLAN | 25 |
| | 7.1 | Statistical Methods | 25 |
| | 7.2 | Sample Size Estimates | 26 |
| | 7.3 | Subject Population(s) for Analysis | 27 |
| | 7.4 | Interim Analysis | 27 |
| | 7.5 | Termination Criteria | 27 |
| | 7.6 | Accountability Procedure | 27 |
| | 7.7 | Deviation Reporting | 27 |
| 8 | DIREC | CT ACCESS TO SOURCE DATA/DOCUMENTATION | 27 |
| 9 | QUAL | ITY CONTROL AND QUALITY ASSURANCE | 27 |
| 10 | ETHIC | CAL CONSIDERATIONS | 28 |



| | | 7 Page |
|----|----------------------------------|----------|
| 11 | DATA HANDLING AND RECORD KEEPING | 28 |
| 12 | FINANCE AND INSURANCE | 29 |



8 | P a g e

#### **List of Abbreviations**

CFR Code of Federal Regulations

CRF Case Report Form

FDA Food and Drug Administration

GCP Good Clinical Practice

IRB Institutional Review Board

EC Ethics Committee

HCP Healthcare Professional

CDC US Center for Disease Control



## 1. Background

#### 1. Overview

During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%). Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2).<sup>3–5</sup> TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro.<sup>6</sup> Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.<sup>7</sup>

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene. 8-10 In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor. 10 Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males. 11

Previously, we have reported the results from two retrospective cohort analysis demonstrating the protective effect of 5-alpha-reductase inhibitors (5ARi) for men with COVID-19.<sup>17</sup> In a study of 77 men hospitalized with COVID-19 we found among men taking 5ARis, 8% were admitted to the ICU compared to 58% of men not taking 5ARis (P = 0.0015). In the cohort, 5ARis were associated with reduced risk for ICU admissions RR 0.14 (95% CI: 0.02–0.94).<sup>17</sup> Similarly, we have demonstrated that the frequency of COVID-19 symptoms was drastically reduced for men using 5ARis in an outpatient setting. A statistically significant (p<0.05) reduction in the frequency of 20 of the 29 clinical symptoms was observed in AGA men using 5ARis compared to AGA men not using 5ARis. For example, 38% and 2% of men presented with low-grade fever, 60% and 6% with dry cough, and 88% and 15% reported anosmia in the non-5ARi and 5ARi groups, respectively.<sup>18</sup>

One limitation of 5ARis is the time course required to achieve systemic DHT reductions. As such, we explored the use of a novel second generation androgen receptor antagonist Proxalutamide as a means for rapid reduction in AR activity. Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the



mechanism that is not present in bicalutamide and enzalutamide. Because of the dual mechanism of action, it is expected to be a more effective and less toxic second-generation anti-androgen drug therapy. Clinical evidence has demonstrated that Proxalutamide lowers AR expression and activity. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells.

In December 2020, we completed a double-blinded, randomized, prospective, investigational study of Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429). The length of the study was 30 days. Proxalutamide was administered 200mg q.d. for 14 days. Men enrolled in the study were 50 years and older. Two hundred and sixty two men completed the study. 134 men were assigned to the Proxalutamide group and 128 men were assigned to the control group. Thirty five subjects were hospitalized in the control group compared to zero in the Proxalutamide group. The proportion of COVID-19 patients hospitalized was significantly different between the Proxalutamide and control arms;  $\chi^2(1) = 42.051$ , p<.0001. The difference in proportions was 27.30% with a 95%CI: [19.79%, 35.59%]. No subject receiving Proxalutamide died compared to 2 (1.56%) in the control group. There were no treatment related adverse event reported during the course of the study.

Based on the results of the Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients study (NCT04446429), the purpose of this study is to assess the efficacy and safety of Proxalutamide as a treatment for hospitalized COVID-19 male patients.

## 1.1. Investigational Drug

#### Proxalutamide (300 mg) q.d.

| Chemical Name | 4-[4,4-dimethyl-3-[6-[3-(2-oxazolyl)propyl]-3-pyridinyl]-5-oxo-2-thioxo-1-imidazolidinyl]-3-fluoro-2-(trifluoromethyl)-benzonitrile |
|---|---|
| CAS Registry No. | 1398046-21-3 |
| Company Code | GT0918 |
| Chemical Structure | N S N N N N N N N N N N N N N N N N N N |
| Molecular Formula | $C_{24}H_{19}F_4N_5O_2S$ |
| Relative Molecular Mass | 517.50 |

Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide.



Because of the dual mechanism of action, it is expected to be a more effective and less toxic second-generation anti-androgen drug therapy. Clinical evidence has demonstrated that Proxalutamide lowers AR expression and activity. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells.

The Proxalutamide tablets (100mg per tablet) will be manufactured by:

TOT BIOPHARM International Company Limited. No. 120 changyang Street, Suzhou Industrial Park, Suzhou City, Jiangsu Province, China

#### 1.1. Pre-Clinical and Prior Clinical Data

#### 1.1.1. Prior Pre-Clinical and Clinical Safety Data

No prior pre-clinical safety data exists as to the use of Proxalutamide for the treatment of COVID-19; however, pre-clinical studies have been conducted in support of the US FDA IND approval of Phase-1 human trials of Proxalutamide in castration resistant prostate cancer. Selected pre-clinical animal studies conducted with Proxalutamide are provided below.

#### Tissue Distribution and Excretion of GT0918 in Rats

The tissue distribution of GT9018 in male SD rats was determined at 0.5, 3 and 12 hours following an oral single administration (20 mg/kg). Proxalutamide was extensively distributed to most of the tissues/organs with high concentrations found in fat tissue and liver, followed by stomach, pancreas and intestine in rats. Proxalutamide distribution was also observed in bone marrow in rats. Peak Proxalutamide concentrations were achieved in most tissues at 3 hours following the administration and a certain degree of elimination was observed in these tissues at 12 hours following the administration.

The excretion profiles (bile, urine and feces) following a single oral dose of Proxalutamide (20 mg/kg) to 6 male SD rats was studied. The data indicated that following a single oral administration of Proxalutamide to rats, the cumulative fractional excretion of Proxalutamide in bile within 36 hours was  $0.010 \pm 0.006\%$ , the cumulative

fractional excretion of Proxalutamide in urine within 72 hours was  $0.014 \pm 0.009\%$  and the cumulative fractional excretion of Proxalutamide in feces within 72 hours was  $10.785 \pm 4.547\%$ . Proxalutamide was mainly excreted in the feces (about 10%) and in trace amounts through bile and urine (0 to 0.1%) in rats.

#### Pharmacokinetic Profiles of Proxalutamide in SD Rats

Pharmacokinetic properties of Proxalutamide were studied in SD rats following single oral dosing at 10, 20, 40 and 80 mg/kg, single IV dosing at 5 mg/kg and repeated PO dosing at 20 mg/kg daily for 8 consecutive days. After single oral dosing, Proxalutamide



reached maximal plasma concentrations in 3 to 5 hours and then decreased with the elimination half-life 2.0 to 2.5 hours. Both AUC and Cmax were proportional to dose. The absolute bioavailability was 74 - 100%. After repeated dosing for 8 days, AUC and Cmax increased about 50% comparing to single dose at the same level, indicating some drug accumulation after repeated dosing.

#### Pharmacokinetic Profiles of Proxalutamide in Beagle Dogs

Pharmacokinetic properties of Proxalutamide were studied in Beagle dogs following single oral dosing at 2, 5 and 10 mg/kg under fasting conditions, single IV dosing at 1 mg/kg, a single oral dosing at 20 mg/kg (with two different API processes) under fed conditions, and repeated PO dosing at 20 mg/kg daily for 7 consecutive days. After single oral dosing, Proxalutamide reached maximal plasma concentrations in 2 to 2.5 hours and then decreased with the elimination half-life 9.5 to 11.8 hours. Both AUC and Cmax were proportional to dose. The absolute bioavailability was 36.5 – 52.5%. Under fed conditions, Cmax markedly decreased about 60% with Tmax increase from 3 hours to 8.3 hours but slightly increased in AUC compared to those respective PK parameters under fasting conditions at the same dose. After repeated dosing for 8 days, AUC and Cmax increased about 70% and 150%, respectively comparing to single dose at the same level, indicating drug accumulation after repeated dosing.

#### 1.1.2 Prior Clinical Safety Data

## Study 1: Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429)

A double-blinded, randomized, prospective, investigational study of Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429) was completed in December 2020. The length of the study was 30 days. Proxalutamide was administered 200mg q.d. for 14 days. Men enrolled in the study were 50 years and older. Two hundred and sixty two men completed the study. 134 men were assigned to the Proxalutamide group and 128 men were assigned to the control group. Thirty five subjects were hospitalized in the control group compared to zero in the Proxalutamide group. The proportion of COVID-19 patients hospitalized was significantly different between the Proxalutamide and control arms;  $\chi 2$  (1) = 42.051, p<.0001. The difference in proportions was 27.30% with a 95%CI: [19.79%, 35.59%]. No subject receiving Proxalutamide died compared to 2 (1.56%) in the control group. There were no treatment related adverse event reported during the course of the study.

#### Study 2: Phase 1 study in 16 males with prostate cancer.

The data from the study was published in a peer review journal. The identifier GT0918 was used to denote Proxalutamide. The abstract from the publication is below:

Abstract Purpose: We conducted preclinical experiments and phase I clinical trial to investigate the safety, pharmacokinetics (PK) and antitumour effects of



GT0918 in castration-resistant prostate cancer (CRPC).

Experimental design: An androgen receptor (AR) competitive binding assay was performed, followed by evaluation of GT0918 on AR protein expression. The efficacy of GT0918 was investigated in a castration-resistant xenograft model. A phase I dose-escalation study of GT0918 in CRPC was also carried out to evaluate its safety, PK and antitumour efficacy. Results: GT0918 was demonstrated to inhibit the binding of androgen to AR more potently than MDV3100, and to effectively reduce the AR protein level. GT0918 inhibited the tran-scriptional activity of wild-type AR and AR with clinically relevant ligand-binding domain mutations. Furthermore, GT0918 significantly inhibited the growth of prostate cancer. A total of 16 patients was treated with GT0918 at five dose levels. Among these 16 patients, 10 and 2 patients, respectively, completed a three-cycle and sixcycle treatment, in which MTD was not reached. All the treatment-related adverse events were grade I, including hypercholesterolemia, hypertriglyceridemia, fatigue and anemia. PK parameters showed that drug exposure increased with dose proportionally from 50 to 300 mg and a saturation was observed between 300mg and 400 mg.

The most significant adverse events from the study are summarized in the following table:

| Table 2 | | | |
|---|---|---|---|
| Most common advers | events of GT0918 | by dose (multiple-dose period | , ≥2 cycles). |

| Adverse event | 50 mg ( | n = 2 | 100 mg | (n=4) | 200 mg (n = 1) | 3) | 300 mg (n = 1) | 3) | 400 mg (n = -1) | Total $(n = 16)$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Drug-<br>related | Drug-<br>irrelative | Drug-<br>related | Drug-<br>irrelative | Drug-related | Drug-<br>irrelative | Drug-related | Drug-irrelative | Drug-related | Drug-<br>irrelative | Drug-<br>related | Drug-<br>irrelative |
| Blood and lymphatic diseases | | | | | | | | | | | | |
| Anaemia | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 |
| Heart diseases | | | | | | | | | | | | |
| Coronary artery disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Visual diseases | | | | | | | | | | | | |
| Eye discomfort | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Gastrointestinal diseases | | | | | | | | | | | | |
| Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |
| Systemic diseases | | | | | | | | | | | | |
| Chest pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| Peripheral oedema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 |
| Abnormal examination results | | | | | | | | | | | | |
| Prolonged coagulation indicators | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| QT interval extension | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| LDH increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| ALP increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| Metabolic and nutritional diseases | | | | | | | | | | | | |
| Hypercholesterolemia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 |
| Malnutrition | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Musculoskeletal and connective<br>tissue diseases | | | | | | | | | | | | |
| Arthralgia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Neurological diseases | | | | | | | | | | | | |
| Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 |
| Urinary diseases | | | | | | | | | | | | |
| Haematuria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Vascular diseases | | | | | | | | | | | | |
| Aortic aneurysm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Hot flushes | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |

LDH, lactate dehydrogenase; ALP, alkaline phosphatase.

Study 3: Phase 1 study conducted in 40 males with prostate cancer.

A summary of the study is provided below:

Demographics: All 40 patients in the Safety Analysis Set were male with the mean age at 70.1 years. Three (7.5%) patients were Hispanic or Latino and 37 (92.5%) were not Hispanic or Latino. Thirty-five (87.5%) patients were white, 4 (10%) were black or



African American and 1 (2.5%) was Asian. Of the 40 patients with mCRPC tumors, all patients (100%) had received at least two lines of hormone therapies, with 11 (27.5%) having 3 lines and 20 (50%) having 4 lines or more. Most patients (70%) had also undergone chemotherapies, with 20 (50%) receiving one line and 8 (20%) receiving 2 or more lines of chemotherapies.

Disposition: The distribution of 40 patients by dose cohort was as follows: 3 at the 50 mg, 6 at the 100 mg, 6 at the 200 mg, 7 at the 300 mg, 7 at the 400 mg, 6 at the 500 mg and 5 at the 600 mg per day dose levels. Of the 40 patients, 1 (2.5%) did not complete 1 cycle, 14 (35%) completed 1 cycle, 10 (25%) completed 2 cycles, 3 (7.5%) completed 3 cycles, 3 (7.5%) completed 4 cycles, 5 (12.5%) completed 5 cycles, and 4 (10%) completed at least 6 cycles of treatment. The primary reason for discontinuation was progressive disease (28/40 patients, 70%). Other discontinuation reasons included the following: unacceptable toxicity or AE (6/40, 15%), withdrawal of consent (4/40, 10%) and patient lost to follow-up (2/40, 5%).

Efficacy: Of the 40 patients, no PSA response with more than 50% reduction from baseline was observed. CR or PR are not required as per phase 1 study data analyses. Treating physicians will do imaging scan to see if patients have with SD allowing for continuing the treatment. The mean number of dosing duration was 12.5 weeks (87.6 days) across all dose cohorts from 50 mg/day to 600 mg/day, and the mean dosing duration for individual dose cohorts ranged from 8.3 weeks (57.7 days) to 15.6 weeks (109.4 days). Patients with treatment duration longer than 22.9 weeks (160 days) were from the following dose cohorts: 1 in the 50 mg/day, 1 in the 100 mg/day, and 2 in the 400 mg/day cohorts. A total of 9 patients had completed between 4 and 6 cycles (28 days per cycle) of treatment, belonging to these dose cohorts: 200 mg/day (1/6), 400 mg/day (4/7), 500 mg/day (2/6), and 600 mg/day (2/5).

Safety: The results from this study showed that the safety profile of GT0918 was generally favorable in patients with mCRPC whose disease progressed after multi-lines of therapies. The mean number of dosing duration was 87.6 days across all dose cohorts from 50 mg/day to 600 mg/day, and the mean dosing duration for individual dose cohorts ranged from 57.7 to 109.4 days. Of the 40 patients, 39 (98%) experienced at least 1 TEAE during the study, with the most frequent AEs being fatigue, nausea, decreased appetite, anemia, weight decrease, diarrhea, constipation, back pain and dizziness. Most of patients reported TEAEs that were considered related to the study drug, with the most common drug-related AEs being fatigue (42.5%), decreased appetite (20%), nausea (15%), dizziness (12.5%), constipation (12.5%), anemia (10%), weight decrease (10%), dysgeusia (10%), and diarrhea (7.5%). Most TEAEs were Grade 1 or 2. Twenty patients across all dose cohorts reported TEAEs of Grade 3 or higher. Each individual TEAE of Grade 3 or higher occurred sporadically in 1 or 2 patients, except for the following: anemia (7/40), fatigue (5/40) and sepsis (3/40). The majority of Grade 3 or higher TEAEs were considered not related to the study drug. Overall, nine patients (9/40, 22.5%) reported at least one SAE. The nine patients were distributed in nearly all dose cohorts except the 100 mg/day cohort. The majority of SAEs were Grade 3 or 4, and two Grade 5 deaths were reported. Both deaths were due to disease progression and they were not related to the study drug. Most SAEs were not drug-related, except for one event of Grade 4 increased creatine phosphokinase (CK). Five patients with SAEs, including sepsis, worsening dehydration, pneumonia and increased CK, were permanently



discontinued from the study. Other drug-related AEs that led to study discontinuation included: fatigue (Grade 3 and Grade 2), anemia (Grade 3) and decreased white blood cell (Grade 3). No DLT was reported in any of the dose cohort. Therefore, MTD was not established in this study. Overall, GT0918 was generally well-tolerated in mCRPC patients.

A summary of AEs are given in the following tables:

Table 12.3 Overview of Treatment-Emergent Adverse Events, Safety Analysis Set

| | | | Esc | alation Col | ort | | | |
|---|---|---|---|---|---|---|---|---|
| | 50 mg/day<br>(N=3)<br>n (%) | 100 mg/day<br>(N=6)<br>n (%) | 200 mg/day<br>(N=6)<br>n (%) | 300 mg/day<br>(N=7)<br>n (%) | 400 mg/day<br>(N=7)<br>n (%) | 500 mg/day<br>(N=6)<br>n (%) | 600 mg/day<br>(N=5)<br>n (%) | Total<br>(N=40)<br>n (%) |
| Adverse Events | 3 (100.0%) | 5 (83.3%) | 6 (100.0%) | 7 (100.0%) | 7 (100.0%) | 6 (100.0%) | 5 (100.0%) | 39 (97.5% |
| Drug-Related Adverse Events | 0 | 3 (50.0%) | 4 (66.7%) | 6 (85.7%) | 6 (85.7%) | 6 (100.0%) | 5 (100.0%) | 30 (75.0% |
| Deaths | 0 | 0 | 0 | 1 (14.3%) | 1 (14.3%) | 0 | 0 | 2 (5.0%) |
| Serious Adverse Events | 1 (33.3%) | 0 | 1 (16.7%) | 2 (28.6%) | 3 (42.9%) | 1 (16.7%) | 1 (20.0%) | 9 (22.5%) |
| Drug-Related Serious Adverse<br>Events | 0 | 0 | 0 | 0 | 0 | 1 (16.7%) | 0 | 1 (2.5%) |
| Adverse Events Leading to<br>Permanent Discontinuation of<br>Study Drug | 0 | 0 | 0 | 3 (42.9%) | 2 (28.6%) | 2 (33.3%) | 2 (40.0%) | 9 (22.5%) |
| Drug-Related Adverse Events<br>Leading to Permanent<br>Discontinuation of Study Drug | 0 | 0 | 0 | 2 (28.6%) | 0 | 2 (33.3%) | 2 (40.0%) | 6 (15.0%) |
| Grade 3 or Higher Treatment-<br>Emergent Adverse Events | 2 (66.7%) | 1 (16.7%) | 3 (50.0%) | 3 (42.9%) | 7 (100.0%) | 2 (33.3%) | 2 (40.0%) | 20 (50.0% |



Table 12.4 Treatment-Emergent Adverse Events by System Organ Class >20%, Safety Analysis Set

| | | | | | | Esc | al | ation Col | OI | t | | | | | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Freferred Term | | GT0918<br>50 mg/day<br>(N=3)<br>n (%) | | GT0918<br>100 mg/day<br>(N=6)<br>n (%) | | GT0918<br>200 mg/day<br>(N=6)<br>n (%) | | GT0918<br>300 mg/day<br>(N=7)<br>n (%) | | GT0918<br>400 mg/day<br>(N=7)<br>n (%) | | GT0918<br>500 mg/day<br>(N=6)<br>n (%) | | GT0918<br>r 600 mg/day<br>(N=5)<br>n (%) | | Total<br>(N=40)<br>n (%) |
| Overall | 3 | (100.0%) | 5 | (83.3%) | 6 | (100.0%) | 7 | (100.0%) | 7 | (100.0%) | 6 | (100.0%) | 5 | (100.0%) | 39 | (97.5% |
| General Disorders And<br>Administration Site Conditions | | | | | | | | | | | | | | (80.0%) | | |
| Fatigue | 2 | (66.7%) | 1 | (16.7%) | 2 | (33.3%) | 4 | (57.1%) | 3 | (42.9%) | 6 | (100.0%) | 3 | (60.0%) | 21 | (52.5% |
| Musculoskeletal And Connective | 2 | (66.7%) | 3 | (50.0%) | 4 | (66.7%) | 5 | (71.4%) | 7 | (100.0%) | 4 | (66.7%) | 1 | (20.0%) | 26 | (65.0% |
| Arthralgia<br>Back Pain | 1 | (33.3%) | 2 | 0<br>(33.3%) | 3 | (50.0%) | | (14.3%)<br>(57.1%) | | (28.6%)<br>(28.6%) | 2 | 0<br>(33.3%) | | 0 | | (25.0% |
| Gastrointestinal Disorders | 1 | (33.3%) | 3 | (50.0%) | 4 | (66.7%) | 3 | (42.9%) | 5 | (71.4%) | 5 | (83.3%) | 4 | (80.0%) | 25 | (62.5% |
| Constipation<br>Diarrhoea | | 0 | | (33.3%) | 1 | Control of the Contro | 1 | | 5 | (28.6%)<br>(71.4%) | 3 | | | 0 | 10 | (25.09 |
| Nausea | 1 | (33.3%) | 1 | (16.7%) | 2 | (33.3%) | 1 | (14.3%) | 4 | (57.1%) | 2 | (33.3%) | 2 | (40.0%) | 13 | (32.5% |
| Nervous System Disorders | 2 | (66.7%) | | | 4 | (66.7%) | | A STATE OF THE PARTY OF THE PAR | | (42.9%) | | | | (60.0%) | | the second second |
| Dizziness | | 0 | 1 | (16.7%) | | 0 | 2 | (28.6%) | 3 | (42.9%) | 2 | (33.3%) | 1 | (20.0%) | 9 | (22.5%) |

Table 12.4 Treatment-emergent Adverse Events by System Organ Class >20%

page 2 of 2

| | | | Esc | alation Col | nort | | | Total |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | GT0918<br>50 mg/day<br>(N=3)<br>n (%) | GT0918<br>100 mg/day<br>(N=6)<br>n (%) | GT0918<br>200 mg/day<br>(N=6)<br>n (%) | GT0918<br>300 mg/day<br>(N=7)<br>n (%) | GT0918<br>400 mg/day<br>(N=7)<br>n (%) | GT0918<br>500 mg/day<br>(N=6)<br>n (%) | GT0918<br>600 mg/day<br>(N=5)<br>n (%) | Total<br>(N=40)<br>n (%) |
| Metabolism And Nutrition<br>Disorders | 1 (33.3%) | 2 (33.3%) | 2 (33.3%) | 4 (57.1%) | 5 (71.4%) | 4 (66.7%) | 3 (60.0%) | 21 (52.5%) |
| Decreased Appetite | 0 | 1 (16.7%) | 1 (16.7%) | 2 (28.6%) | 3 (42.9%) | 3 (50.0%) | 2 (40.0%) | 12 (30.0%) |
| Investigations | 1 (33.3%) | 1 (16.7%) | 1 (16.7%) | 4 (57.1%) | 3 (42.9%) | 4 (66.7%) | 1 (20.0%) | 15 (37.5%) |
| Weight Decreased | 1 (33.3%) | 0 | 1 (16.7%) | 1 (14.3%) | 3 (42.9%) | 3 (50.0%) | 1 (20.0%) | 10 (25.0%) |
| Respiratory, Thoracic And<br>Mediastinal Disorders | 2 (66.7%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 4 (57.1%) | 1 (16.7%) | 2 (40.0%) | 15 (37.5%) |
| Blood And Lymphatic System<br>Disorders | 1 (33.3%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 4 (57.1%) | 1 (16.7%) | 1 (20.0%) | 13 (32.5% |
| Anaemia | 1 (33.3%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 3 (42.9%) | 1 (16.7%) | 0 | 11 (27.5%) |
| Infections And Infestations | 2 (66.7%) | 0 | 0 | 2 (28.6%) | 4 (57.1%) | 0 | 3 (60.0%) | 11 (27.5% |
| Vascular Disorders | 0 | 3 (50.0%) | 1 (16.7%) | 2 (28.6%) | 4 (57.1%) | 0 | 1 (20.0%) | 11 (27.5%) |
| Renal And Urinary Disorders | 1 (33.3%) | 0 | 2 (33.3%) | 3 (42.9%) | 1 (14.3%) | 1 (16.7%) | 0 | 8 (20.0%) |
| Cardiac Disorders | 1 (33.3%) | 0 | 0 | 2 (28 6%) | 3 (42 99) | 1 (16 79) | 1 (20.0%) | 8 (20.0%) |

Study 4: Phase II dose escalating study of Proxalutamide (100-300 mg) in 108 patients with prostate cancer.

A table of adverse events observed in the trial are described below.


This material is the property of the Applied Biology Inc. Do not disclose or use except as authorized.



| PT name | 100 mg<br>(N=37)% | 200 mg<br>(N=35)% | 300 mg<br>(N=36)% | Total<br>(N=108)% | P |
|---|---|---|---|---|---|
| Asthenia/ fatigue | 2 (5.4) | 7 (20.0) | 14 (38.9 | 23 (21.3) | < 0.05 |
| Aspartate aminotransferase | 5 (13.5) | 5 (14.3) | 6 (16.7) | 16 (14.8) | >0.05 |
| Anaemia | 3 (8.1) | 7 (20.0) | 6 (16.7) | 16 (14.8) | >0.05 |
| Alanine aminotransferase increased | 6 (16.2) | 4 (11.4) | 4 (11.1) | 14 (13.0) | >0.05 |
| Decreased appetite | 3 (8.1) | 3 (8.6) | 8 (22.2) | 14 (13.0) | >0.05 |
| White blood cell count decreased | 2 (5.4) | 5 (14.3) | 6 (16.7) | 13 (12.0) | >0.05 |
| Proteinuria | 4 (10.8) | 4 (11.4) | 5 (13.9) | 13 (12.0) | >0.05 |
| Constipation | 1 (2.7) | 3 (8.6) | 6 (16.7) | 10 (9.3) | >0.05 |
| Oedema peripheral | 1 (2.7) | 4 (11.4) | 3 (8.3) | 8 (7.4) | >0.05 |
| Blood fibrinogen increased | 2 (5.4) | 2 (5.7) | 3 (8.3) | 7 (6.5) | >0.05 |
| Blood triglycerides increased | 5 (13.5) | 2 (5.7) | 0 | 7 (6.5) | >0.05 |
| Neutrophil count decreased | 0 | 4 (11.4) | 3 (8.3) | 7 (6.5) | >0.05 |
| Weight decreased | 1 (2.7) | 2 (5.7) | 4 (11.1) | 7 (6.5) | >0.05 |
| Hypertriglyceridaemia | 1 (2.7) | 3 (8.6) | 3 (8.3) | 7 (6.5) | >0.05 |
| Nausea | 1 (2.7) | 0 | 6 (16.7) | 7 (6.5) | < 0.05 |
| Supraventricular extrasystoles | 1 (2.7) | 3 (8.6) | 2 (5.6) | 6 (5.6) | >0.05 |
| Haematuria | 2 (5.4) | 3 (8.6) | 1 (2.8) | 6 (5.6) | >0.05 |
| Platelet count decreased | 2 (5.4) | 1 (2.9) | 2 (5.6) | 5 (4.6) | >0.05 |

#### **Drug Interactions**

Inhibition Potential Assessment of Proxalutamide on Cytochrome P450 Enzymes in Pooled Human Liver Microsomes

The inhibition of human liver CYPs: CYP1A2, CYP2C9, CYP2C19, CYP2D6, CYP2E1 and CYP3A4/5, was assessed with Proxalutamide at concentrations of 0.2, 0.8, 2, 10, 50, 100 and 200  $\mu$ M. The metabolite formation from CYP catalyzed probe substrate metabolism was analyzed with LC-MS/MS. The results showed that Proxalutamide showed no significant inhibition on CYP1A2 and CYP2E1, weak inhibition on CYP2D6, CYP2C9, CYP2C19 and CYP3A (midazolam), but marked inhibition on CYP3A4 (testosterone).

The results indicate that there is an inhibitory effect of Proxalutamide on CYP3A4 in vitro and the corresponding in vivo drug interaction potential needs to be further investigated.

\*No interaction has been reported between Proxalutamide, nitazoxanide, and azithromycin.



| <b>Table 1.2.3:</b> | Inhibitory Effect of Proxalutamide on CYP450 Enzymes | | | |
|---|---|---|---|---|
| CYP450s | Probe substrate | Characterized<br>Metabolic<br>Pathway | Characterized Metabolite | IC <sub>50</sub> (MM) |
| CYP1A2 | Phenacetin | Deethylation | Acetaminophen | >200 |
| CYP2C9 | Tolbutamide | Hydroxylation | 4-Hydroxy-Tolbutamide | 8 |
| CYP2C19 | Omeprazole | Hydroxylation | 5-Hydroxy- Omeprazole | 8 |
| CYP2D6 | Dextromethorphan | Demethylation | Dextrorphan | 5 |
| CYP3A4 | Midazolam | Hydroxylation | 1-Hydroxy-Midazolam | 56 |
| CYP3A4 | Testosterone | Hydroxylation | 6β-Testosterone | 1 |
| CYP2E1 | Chlorzoxazone | Hydroxylation | 6-Hydroxy-Chlorzoxazone | >200 |

<u>Evaluation of Cytochrome P450 Induction Potential of Proxalutamide in Human Hepatocytes</u>

Proxalutamide was evaluated for induction of drug metabolizing enzymes in primary human hepatocytes. No inductive effects on CYP1A2 and CYP3A4 were observed in the level of enzymatic activity.

Table 10: Effect of Proxalutamide on the Enzyme Activity of CYP1A2

| | Activity | of CYP1A | 2 (%) | Mean | SD | Activity compared to positive control (%) |
|---|---|---|---|---|---|---|
| Negative control | 109 | 82.4 | 108 | 100 | 15.2 | NA |
| Positive control | 1174 | 1246 | 1207 | 1209 | 36.3 | 100 |
| Proxalutamide 1 µM | 98.9 | 98.2 | 95.6 | 97.6 | 1.74 | <40 |
| Proxalutamide 10 µM | 92.3 | 98.9 | 99.6 | 96.9 | 4.01 | <40 |

| Table 11: Effect of PROXALUTAMIDE on the Enzyme Activity of CYP3A4 | | | | | | |
|---|---|---|---|---|---|---|
| Control | Activit | y of CYP3A | 4(%) | Mean | SD | Activity compared to positive control (%) |
| Negative control | 97.3 | 103 | 99.6 | 100 | 2.97 | NA |
| Positive control | 805 | 976 | 825 | 869 | 93.4 | 100 |
| Proxalutamide 1 µM | 24.2 | 26.0 | 27.7 | 26.0 | 1.73 | <40 |
| Proxalutamide 10μM | 19.7 | 21.3 | 19.4 | 20.2 | 1.05 | <40 |

## **Specific Populations**



#### **Pediatric**

Proxalutamide pharmacokinetics have not been investigated in subjects younger than 18 years.

#### Geriatric

No dose adjustment is necessary in the elderly. The pharmacokinetics and pharmacodynamics of Proxalutamide were evaluated in 40 patients with an average age of 70.1 (Study 2, Section 1.1.2.4.).

#### Gender

Proxalutamide is not indicated for use in women. The palnned interventional study will be conducted in men only.

#### Race

The effect of race on Proxalutamide pharmacokinetics has not been studied.

#### <u>Renal Impairment</u>

The effect of renal impairment on Proxalutamide pharmacokinetics has not been studied.

#### **Hepatic Impairment**

The effect of hepatic impairment on Proxalutamide pharmacokinetics has not been studied.

#### 1.1.3 Prior Pre-clinical Efficacy Data

No prior pre-clinical data exists as to the use of Proxalutamide as a treatment for COVID-19.; however, two studies highlight the possible benefit of the dual anti-androgen activity of Proxalutamide.

#### Proxalutamide inhibition of androgen binding to AR and AR protein expression

A study by Zhou et al<sup>19</sup> reported that: "GT0918 inhibited the binding of androgen to AR in a dose-dependent manner, and the Ki value of GT0918 (1.4 x 10<sup>-8</sup> M) in binding to AR was 3.4-fold lower than that of MDV3100 (4.8 x 10<sup>-8</sup> M) (Fig. 1A). It indicated that GT0918 was more potent than MDV3100 in inhibiting the binding of androgen to AR." Additionally, in cultures of C4-2B cells, "the protein expression of AR was significantly reduced by GT0918". Data depicting the inhibition androgen binding to AR and the reduced AR protein expression in C4-2B cells is shown below:





Fig. 1. GT0918 effectively decreases androgen binding to AR. (A) IC<sub>50</sub> values for GT0918 and MDV3100 in inhibiting androgen from binding to AR. (B) GT0918 reduces the protein expression of AR in C4-2B cells.

### Proxalutamide suppression ACE2 and TMPRSS2 in A549 lung cells

A study by Wu et al <sup>20</sup> reported that "In LNCaP and A549 cells, we showed that androgen induced the ACE2 and TMPRSS2 expression, and GT0918 could suppress the ACE2 and TMPRSS2 expression". The data from the study is depicted in the figure below.



#### 1.1.4 Prior Clinical Efficacy Data



## Study 1: Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429)

Proxalutimede has been studied in a prospective clinical trial as a treatment for non-hospitalized COVID-19 male patients. A summary of the study and the results are as follows:

Objective: To determine if the anti-androgen Proxalutamide is an effective treatment for men not-hospitalized due to COVID-19 disease (based on assessment of the clinical status on an 8 point ordinal scale: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities) Design: A double-blinded, randomized, prospective, investigational study of Proxalutamide as a treatment for non-hospitalized COVID-19 male patients (inclusion ordinal scale <3).

**Setting:** Outpatient centers (Brasilia, Brazil) from July 15 to December 24, 2020. Participants: Men not hospitalized due to COVID-19 disease (inclusion ordinal scale <3) **Interventions:** Proxalutamide 200mg/day, or standard of care for 14 days.

Main Outcome and Measures: Percentage of subjects hospitalized due to COVID-19 [Time Frame: 30 days]

**Results:** A total of 268 men were included and completed the trial; 134 men were randomized to the Proxalutamide group, and 128 men were randomized to the control group. Data is summarized in Table 1.4.1. A statistically significant difference (p<0.001) in the percentage of subjects hospitalized due to COVID-19 was observed in men taking Proxalutamide compared to the standard of care. The percentage of men hospitalized were 2.2% and 26% in the Proxalutamide and control groups, respectively. No subject receiving Proxalutamide died versus 2 (1.56%) in the control group.

**Conclusions and Relevance:** Non-hospitalized COVID-19 male patients (inclusion ordinal scale <3) treated with Proxalutamide, had significantly reduced rate of hospitalization compared to men not receiving Proxalutamide.

Trial Registration: NCT04446429

| | Control | Proxalutamide |
|------------------|---------|---------------|
| Not Hospitalized | 99 | 131 |
| Hospitalized | 35 | 3 |
| Total | 134 | 134 |

Table 1.4.1 Clinical outcomes of COVID-19 male patients treated with Proxalutamide compared to standard of care.

#### 1.1.5 Justification for Dosage



According to a phase I study of Proxalutamide conducted by Zhou et al<sup>19</sup> PK parameters showed that drug exposure increased with dose proportionally from 50 to 300 mg and a saturation was observed between 300mg and 400 mg.

Further, the research team conducting the NCT04446429 study had previously administered to five COVID-19 male patients Proxalutamide at dosages as high as 400mg q.d. These patients did not qualify to be enrolled in the study due to age <50. In the assessment of the research team, these patients were at an imminent threat of hospitalization due to COVID-19. All patients have exhibited shortness of breath, coughing and oxygen saturation <=93%. A marked improvement in symptoms was observed 24 hours following administration of 400mg Proxalutamide. None of the imminent were subsequently hospitalized. No treatment related adverse events were observed.

As such, we believe that Proxalutamide 300mg q.d.is likely to provide efficacy in the treatment of hospitalized COVID-19 male patients without increasing the rate of treatment related adverse events (none observed in NCT04446429)

#### 1.1.6 Other Data

The PI has not identified any additional data related to the safety or efficacy of this study.

## 1.2. Risks/Benefits

This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study to assess the efficacy of Proxalutamide as a treatment for hospitalized COVID-19 male patients; therefore, we assess below the risks/benefits for the proposed study.

#### **Benefit(s) of the Proposed Clinical Study**

To-date no therapy for hospitalized COVID-19 patients has demonstrated significant clinical benefit. Proxalutamide demonstrated clinical efficacy in non-hospitalized COVID-19 male patients (NCT04446429). As such, subjects enrolled in this study could potentially benefit from reduced hospitalization time as well as lower risk of experiencing progressively more severe COVID-19 related symptoms. In addition, if Proxalutamide demonstrates clinical efficacy in this study, it is likely to improve the standard of care for hospitalized COVID-19 male patients world-wide.

#### Risk(s) of the Proposed Clinical Study

Treatment with any drug carries risk. Treatment with Proxalutamide caries the risk of the adverse events reported in Phase I clinical trials with Proxalutamide; however, due to the short treatment duration of 14 days, we believe the risk of serious adverse events is lower than described in Phase I studies. Further, during 14 days of dosing 134 subjects with 200mg q.d. of Proxulatimde no drug related adverse events were observed.



#### 1.3. Trial Conduct

This study will be conducted in compliance with the protocol approved by the Institutional Review Board (Ethics Committee), and according to Good Clinical Practice standards. No deviation from the protocol will be implemented without the prior review and approval of the IRB (EC) except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the IRB (EC) as soon as possible.

## 1.4. Population

This is a multi-center study to be conducted at hospital sites. This exact protocol will be followed. There will be one or more PIs. The study will be approved by each hospital's Ethics Committee.

The population for this study will be hospitalized COVID-19 male patients 18 years or older of any ethnicity. Approximately, 300 male subjects who meet all the eligibility criteria will be enrolled. The estimated time from screening to end of the study for each subject is approximately 14 days.

#### 1.5. Literature

- 1. Guan W-J, Ni Z-Y, Hu Y, et al. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. February 2020:NEJMoa2002032. doi:10.1056/NEJMoa2002032
- 2. Goren A, Mc Coy J, Wambier CG, et al. WHAT DOES ANDROGENETIC ALOPECIA HAVE TO DO WITH COVID-19? AN INSIGHT INTO A POTENTIAL NEW THERAPY. Dermatol Ther. April 2020:e13365. doi:10.1111/dth.13365
- 3. Shieh WJ, Hsiao CH, Paddock CD, et al. Immunohistochemical, in situ hybridization, and ultrastructural localization of SARS-associated coronavirus in lung of a fatal case of severe acute respiratory syndrome in Taiwan. Hum Pathol. 2005. doi:10.1016/j.humpath.2004.11.006
- 4. Hoffmann M, Kleine-Weber H, Schroeder S, et al. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. March 2020:1-10. doi:10.1016/j.cell.2020.02.052
- 5. Glowacka I, Bertram S, Muller MA, et al. Evidence that TMPRSS2 Activates the Severe Acute Respiratory Syndrome Coronavirus Spike Protein for Membrane Fusion and Reduces Viral Control by the Humoral Immune Response. J Virol. 2011. doi:10.1128/jvi.02232-10
- 6. Heurich A, Hofmann-Winkler H, Gierer S, Liepold T, Jahn O, Pohlmann S. TMPRSS2 and ADAM17 Cleave ACE2 Differentially and Only Proteolysis by TMPRSS2 Augments Entry Driven by the Severe Acute Respiratory Syndrome Coronavirus Spike Protein. J Virol. 2014;88(2):1293-1307. doi:10.1128/JVI.02202-13
- 7. Limburg H, Harbig A, Bestle D, et al. TMPRSS2 Is the Major Activating Protease of Influenza A Virus in Primary Human Airway Cells and Influenza B Virus in Human Type II Pneumocytes. Schultz-Cherry S, ed. J Virol. 2019;93(21). doi:10.1128/JVI.00649-19
- 8. Lucas JM, Heinlein C, Kim T, et al. The Androgen-Regulated Protease TMPRSS2 Activates a Proteolytic Cascade Involving Components of the Tumor Microenvironment and Promotes Prostate Cancer Metastasis. Cancer Discov. 2014;4(11):1310-1325. doi:10.1158/2159-8290.CD-13-1010



- 9. National Institutes of Health. TMPRSS2 transmembrane serine protease 2 [ Homo sapiens (human) ] Gene ID: 7113. Gene ID: 7113, updated on 13-Mar-2020. https://www.ncbi.nlm.nih.gov/gene/7113. Published 2020. Accessed April 2, 2020. 10. Lin B, Ferguson C, White JT, et al. Prostate-localized and androgen-regulated expression of the membrane- bound serine protease TMPRSS2. Cancer Res. 1999.
- 11. Dalpiaz PLM, Lamas AZ, Caliman IF, et al. Sex Hormones Promote Opposite Effects on ACE and ACE2 Activity, Hypertrophy and Cardiac Contractility in Spontaneously Hypertensive Rats. Bader M, ed. PLoS One. 2015;10(5):e0127515. doi:10.1371/journal.pone.0127515
- 12. Gan DCC, Sinclair RD. Prevalence of male and female pattern hair loss in Maryborough. J Investig Dermatol Symp Proc. 2005;10(3):184-189. doi:10.1111/j.1087-0024.2005.10102.x 13. Goren et al. A PRELIMINARY OBSERVATION: MALE PATTERN HAIR LOSS AMONG HOSPITALIZED COVID-19 PATIENTS IN SPAIN A POTENTIAL CLUE TO THE ROLE OF ANDROGENS IN COVID-19 SEVERITY. J. Cos. Derm (accepted April 2020)
- 14. Severi G, Sinclair R, Hopper JL, English DR, McCredie MR, Boyle P, Giles GG. Androgenetic alopecia in men aged 40-69 years: prevalence and risk factors. Br J Dermatol. 2003; 149(6): 1207-1213.
- 15. Hamilton JB. Patterned loss of hair in man: Types and incidence. Ann N Y Acad Sci. 1951;53:708–728.
- 16. Montopoli M, Zumerle S, Vettor R, Rugge M, Zorzi M, Catapano CV, Carbone GM, Cavalli A, Pagano F, Ragazzi E, Prayer-Galetti T, Alimonti A, Androgen-deprivation therapies for prostate cancer and risk of infection by SARS-CoV-2: a population-based study (n=4532), Annals of Oncology (2020), doi: <a href="https://doi.org/10.1016/j.annonc.2020.04.479">https://doi.org/10.1016/j.annonc.2020.04.479</a>
  17. Goren A, Wambier CG, Herrera S, McCoy J, Vaño-Galván S, Gioia F, Comeche B, Ron R, Serrano-Villar S, Ramos PM, Cadegiani FA, Kovacevic M, Tosti A, Shapiro J, Sinclair R. Anti-androgens may protect against severe COVID-19 outcomes: results from a prospective cohort study of 77 hospitalized men. J Eur Acad Dermatol Venereol. 2020 Sep 25:10.1111/jdv.16953. doi: 10.1111/jdv.16953. Epub ahead of print. PMID: 32977363; PMCID: PMC7536996.
- 18. McCoy J, Cadegiani FA, Wambier CG, Herrera S, Vaño-Galván S, Mesinkovska NA, Ramos PM, Shapiro J, Sinclair R, Tosti A, Goren A. 5-Alpha-Reductase Inhibitors are Associated with Reduced Frequency of COVID-19 Symptoms in Males with Androgenetic Alopecia. J Eur Acad Dermatol Venereol. 2020 Nov 2. doi: 10.1111/jdv.17021. Epub ahead of print. PMID: 33135263.
- 19. Zhou T, Xu W, Zhang W, Sun Y, Yan H, Gao X, Wang F, Zhou Q, Hou J, Ren S, Yang Q, Yang B, Xu C, Zhou Q, Wang M, Chen C, Sun Y. Preclinical profile and phase I clinical trial of a novel androgen receptor antagonist GT0918 in castration-resistant prostate cancer. Eur J Cancer. 2020 Jul;134:29-40. doi: 10.1016/j.ejca.2020.04.013. Epub 2020 May 24. PMID: 32460179.
- 20. Wu, Siqi and Miao, Liyan and Zhou, Qianxiang and Gao, Chang and Liu, Jialin and Zhan, Qingyuan and Guo, Binbin and Li, Fang and Wang, Yirong and Xu, Hongyang and Yan, Honghua and Wu, Rui and Zhang, Shenghua and Zheng, Jiangnan and Yang, Jianfei and Wang, Shanshan and Yu, Wenkui and Niu, Haitao and Li, Fengyuan and Yang, Ling and Huang, Jianan and Lu, Xiaoting and Chen, Jiahao and Tong, Youzhi and Ma, Liandong and Zhou, Yifeng and Guo, Qiang, Suppression of Androgen Receptor (AR)-ACE2/TMPRSS2



Axis by AR Antagonists May Be Therapeutically Beneficial for Male COVID-19 Patients (April 20, 2020). Available at

SSRN: <a href="https://ssrn.com/abstract=3580526">https://ssrn.com/abstract=3580526</a> or <a href="https://dx.doi.org/10.2139/ssrn.3580526">https://dx.doi.org/10.2139/ssrn.3580526</a>

## 2. Trial Objectives

The primary purpose of this study is to evaluate the efficacy of Proxalutamide as a treatment for hospitalized COVID-19 male patients.

## 3. Trial Design

#### 3.1 Primary Study Endpoints/Secondary Endpoints

#### **Primary Outcome Measure:**

1. Treatment efficacy of Proxalutamide relative to placebo arm as assessed by the COVID-19 ordinal scale (defined in Section 5.1) [Time Frame: Day 14]

#### **Secondary Outcome Measures:**

- Mean change in clinical symptoms assessed by the COVID-19 ordinal scale (defined in Section 5.1) [Time Frame: Day 1, 14, 28]
   A negative change indicates improvement in symptoms and a positive change indicates worsening symptoms
- 2. Time to recovery [Time Frame: Day 1 through Day 28]
  Recovery is defined as the first day on which the subject satisfies one of the following two categories from the ordinal scale (defined in Section 5.1): 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
- 3. Treatment efficacy of Proxalutamide relative to placebo arm as assessed by the COVID-19 ordinal scale (defined in Section 5.1) [Time Frame: Day 28]

## 3.2 Study Design/Type

This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study. The study will have 2 arms:

Arm 1: Subjects administered Nitazoxanide 500 mg b.i.d for 5 days + azithromycin 500mg q.d for 5 days + Proxalutamide 300mg q.d for 14 days

Arm 2: Subjects administered Nitazoxanide 500 mg b.i.d for 5 days + azithromycin 500mg q.d for 5 days + Proxalutamide placebo 300mg q.d for 14 days



#### **Study Environment:**

This is a multi-center study to be conducted at multiple hospitals (the sites). This exact protocol will be followed during the study. There will be one or more PIs. The study will be approved by the appropriate Ethics Committees (IRBs). Data collection will be performed at each site by study personnel under the supervision of the PI.

#### **Study Design:**

#### Phase I: Enrollment (within 24 hours of admission to hospital):

- 1. Each subject will be evaluated for the inclusion and exclusion criteria
- 2. Each subject will undergo a physical examination
- 3. Each subject (or legally authorized representative) will complete and sign the Informed Consent Form
- 4. Each subject will be assigned a subject study number
- 5. Each subject will be randomly assigned to an Arm (Section 3.3)
- 6. Based on the Arm assignment, each subject will be administered the intervention
- 7. All information will be recorded in the appropriate CRFs

#### Phase II: Outcome Assessment at Site (days 1-14):

- 1. Each subject will be evaluated daily by the PI for the outcomes of this study
- 2. Based on the Arm assignment, each subject will be administered the intervention
- 3. The PI will assess each subject for any treatment related adverse events
- 4. All information will be recorded in the appropriate CRFs

#### 3.3 Randomization

Subjects will be randomized into 1 of 2 arms each will receive an interventional treatment.

Arm 1: Subjects administered Nitazoxanide 500 mg b.i.d for 5 days + azithromycin 500mg q.d for 5 days + Proxalutamide 300mg q.d for 14 days



Arm 2: Subjects administered Nitazoxanide 500 mg b.i.d for 5 days + azithromycin 500mg q.d for 5 days + Proxalutamide placebo 300mg q.d for 14 days

During the enrollment phase (admission to hospital), each subject will be assigned a subject study number. The first subject will be assigned the number 001 and each subject thereafter will be assigned a consecutive number i.e., 002, 003, etc. The randomization plan is based on a 1:1 ratio for each arm. Since the study is double-blinded, the following randomization schedule will be used but the identification of the Arm assignment will be known only to the sponsor:

```
Subjects 001-020 will be assigned to Arm 1
Subjects 021-040 will be assigned to Arm 2
Subjects 041-060 will be assigned to Arm 1
Subjects 061-080 will be assigned to Arm 2
Subjects 081-100 will be assigned to Arm 1
Subjects 101-120 will be assigned to Arm 2
etc......
```

#### 3.4 Records

Each subject will be assigned a number. The numbers will be consecutive starting at 001.

A record will be created for each subject. Each record will contain a medical history, and the subject's efficacy parameters copied from the subject's charts and documented in the appropriate CRF.

The subjects' records will be stored and handled in the same manner as the PI's other clinical study patients' records are stored i.e., in a locked research storage area.

No other data will be recorded. No personal information will be kept outside the study site.

Data compiled at the end of the study will not include any information that can be used to identify individuals.

#### 3.5 Duration

The duration of the study is 28 days. There will be no study related follow-up treatment.

#### 3.6 Discontinuation

In the event that a subject reports any drug related adverse event (not ARDS symptom) we will discontinue the study for that particular subject.

In the event a subject in any arm experiences a serious adverse event defined as death not due to respiratory failure (presents with clear lung CT and no ARDS symptoms) the study will be discontinued. The reminder of the study shall continue.

## 3.7 Product Accountability

All interventional treatments for this study will be stored and monitored according to each



hospital standard protocol.

## 3.8 Data Identification

The subject records kept by the PI will be stored and handled in the same manner as the PI's other clinical research subject records. Only authorized personnel named in this study, or medical professional retained by the PI in case of an adverse event, will have access to the subject records.

No other data will be recorded. No personal information will be kept outside the study site.

Data compiled at the end of the study will not include any information that can be used to identify individuals.

## 4. Selection and Withdrawal of Subjects

#### 4.1 Inclusion Criteria

- 1. Admitted to the hospital with symptoms of COVID-19
- 2. Male age  $\geq$ 18 years old
- 3. Laboratory confirmed positive SARS-CoV-2 rtPCR test in the past 7 days
- 4. Clinical status on the COVID-19 Ordinal Scale (defined in Section 5.1) of 3, 4 or 5
- 5. Coagulation: INR  $\leq 1.5 \times ULN$ , and APTT  $\leq 1.5 \times ULN$
- 6. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
- 7. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

## 4.2 Exclusion Criteria

- 1. Subject enrolled in a study to investigate a treatment for COVID-19
- 2. Requires mechanical ventilation
- 3. Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc...
- 4. Patients who are allergic to the investigational product or similar drugs (or any excipients);
- 5. Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
- 6. Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
  - 7. Subjects with uncontrolled medical conditions that could compromise participation in the study(e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
  - 8. Known diagnosis of human immunodeficiency virus(HIV), hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory)
  - 9. Subject likely to transfer to another hospital within the next 14 days



10. Subject (or legally authorized representative) not willing or unable to provide informed consent

#### 4.3 Subject Withdrawal

Subjects may withdraw at any time for any reason. In the event the principal investigator or the site monitor believes a subject is at risk of injury the subject will be withdrawn from the study and:

- (a) If the subject has not completed the study
- (b) The subject will be replaced with another subject
- (c) The PI will follow-up with the subject every day for 14 days
- (d) The information will be reported in the appropriate CRF

## 4.4 Treatment of Subjects

Once enrolled in the study, the PI or the PI's assistant will administer the assigned treatment on a daily basis at the hospital site.

#### 4.5 Medication

Proxalutamide showed no significant inhibition on CYP1A2 and CYP2E1, weak inhibition on CYP2D6, CYP2C9, CYP2C19 and CYP3A (midazolam), but obvious inhibition on CYP3A4 (testosterone). Potential inducer on CYP3A4 at a concentration of 10μM. No inductive effects on CYP1A2 and CYP2B6 were observed in the level of enzymatic activity. Co-administration of strong/moderate CYP3A4 inducer, strong/moderate CYP3A4 inhibitor, sensitive CYP3A4/ CYP2D6 substrates and narrow therapeutic index with Proxalutamide should be used cautiously (See Appendix 1).

Note: No interaction has been reported between Proxalutamide, Nitazoxanide, and azithromycin.

Therapy prior to enrollment with any other treatment for COVID-19 or the SARS-CoV-2 infection are permitted but must be discontinued on enrollment. There is no waiting period between discontinuation of these treatments and administration of the study intervention; however, these prior treatments and their end date should be documented in the Concomitant Medication CRF.

## 4.6 Monitoring for subject compliance

The PI will monitor each subject's chart to assure daily administration of the treatment by the study staff.



## 5 Assessment of Efficacy

## 5.1 Efficacy Parameters

The following efficacy parameters will be assessed and recorded in the CRF.

#### **I. COVID-19 Ordinal Scale:**

The ordinal scale is an assessment of the clinical status of each subject. The scale is defined as follows:

- 8. Death:
- 7. Hospitalized, on invasive mechanical ventilation or ECMO;
- 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
- 5. Hospitalized, requiring supplemental oxygen;
- 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise;
- 3. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care;
- 2. Not hospitalized, limitation on activities;
- 1. Not hospitalized, no limitations on activities

#### II. Time to Recovery:

Time to recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale (defined in Section 5.1): 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; or 1) Not hospitalized, no limitations on activities.

## 5.2 Method and Timing

For each study day while the subject is hospitalized, the PI will record the clinical assessment on an 8- point ordinal scale as follows:

- Day 1 The clinical assessment at the time of enrollment.
- Day 2 The most severe clinical assessment occurring any time between enrollment and midnight the day following enrollment.
- Day 3-14 (or until discharged) The most severe assessment occurring from midnight to midnight of the prior day (e.g., the value recorded on Day 3 will be the most severe outcome that occurred on Day 2).

If the subject is no longer hospitalized at day 14, a clinical assessment will be made by an inperson or phone visit.



## **6** Assessment of Safety

## 6.1 Safety Parameters

Safety parameters will be assessed as follows:

#### I. Physical Examination:

The PI will conduct a thorough physical examination during screening. The assessment will be recorded in the appropriate CRF.

## **II. Clinical Laboratory Evaluations:**

The following tests will be conducted: WBC, differential, Hgb, PLT, creatinine, glucose, total bilirubin, AST, ALT and coagulation PT.

#### **III. Adverse Events:**

Safety will be assessed by summarizing the incidence and type of Adverse Events in a CRF form.

## 6.2 Method and Timing

The assessments, as described in section 6.1, will occur as follows:

#### **I. Physical Examination**

The assessment will occur at screening. The information will be recorded in the appropriate CRF.

#### **II. Clinical Laboratory Evaluations:**

The assessment will occur upon admission to the hospital as well as at day 14. Additional laboratory tests or timing may be ordered as deemed necessary by the PI.

#### **III. Adverse Events:**

Adverse events will be assessed daily during the 14-day duration of the trial. The information will be recorded in the appropriate CRF.

The methods employed for completing assessments are described in section 6.1

## 6.3 Adverse Event Reporting

We will comply with any EC/IRB and/or FDA requirements for adverse events reporting.

The following events will be reported within 10 days (unless otherwise indicated below):

• Any serious event (including on-site and off-site adverse events, injuries, side effects, deaths or other problems) which in the opinion of the local investigator was unanticipated, involved risk to subjects or others, and was possibly related to the research procedures will be reported within 24 hours.



- Any serious accidental or unintentional change to the IRB-approved protocol that involves risk or has the potential to recur will be reported within 24 hours.
- Any deviation from the protocol taken without prior IRB review to eliminate apparent immediate hazard to a research subject.
- Any publication in the literature, safety monitoring report (including Data and Safety Monitoring Reports), interim result or other finding that indicates an unexpected change to the risk/benefit ratio of the research.
- Any breach in confidentiality that may involve risk to the subject or others.
- Any complaint of a subject that indicates an unanticipated risk or that cannot be resolved by the research staff will be reported within 24 hours.
- Any other serious and possibly related event which in the opinion of the investigator constitutes an unanticipated risk will be reported within 24 hours.

In the event of any adverse event during or after the trial we will keep records of such events in the appropriate CRFs, report to the IRB/FDA and any treating physician if necessary.

## 6.4 Definitions

- Unanticipated (unexpected) problems/events are those that are *not* already described as potential risks in the consent form, *not* listed in the Investigator's Brochure or *not* part of an underlying disease. Anticipated (expected) problems/events do NOT meet the IRB's definition of UPIRTSO.
- **Serious** problems/events are those which in the opinion of the local investigator involve risk to subjects or others. Examples may include death, hospitalization, disability as well as breach of confidentiality. **Non-serious** problems/events do NOT meet the IRB's definition of UPIRTSO.
- Problems/events that are unanticipated and serious should be reported to the IRB within 10 working days *only* if in the opinion of the local investigator they are possibly, probably or definitely **related** to the research procedures. Those serious, unanticipated problems/events that the local investigator deems unlikely or **not related** do NOT meet the IRB's definition of UPIRTSO.
- Follow-up reports on previous events should be reported as UPIRTSOs if the initial event itself met the IRB's definition of UPIRTSO **AND** in the local investigator's judgment, this follow-up report adds value to the initial report.
- Reports of off-site events on studies that are now closed at this site should be reported as UPIRTSOs if the event meets the IRB's definition of UPIRTSO AND in the local investigator's judgment, this event may affect risk to subjects who have completed the study.
- For reports involving blinded study drug, the assessment of relatedness will often be "at least possibly related" as relatedness cannot always be ruled out. If there are numerous reports on the same blinded drug and these reports all meet the 3 criteria for UPIRTSO, they may be reported on one UPIRTSO form with an accompanying table/spreadsheet. A



narrative regarding whether risk is altered or subjects should be notified may be provided for each group of similar events.

## 6.5 Adverse Event Follow-up

Follow-up daily for the first 30 days following drug related adverse event; thereafter, every 7 days up to an additional 90 days.

#### 7 Statistical Plan

#### 7.1 Statistical Methods

#### **I. General Principles:**

- Double-blinded, placebo controlled randomized interventional study with a two-sided type I error rate of 0.05.
- Continuous variables will be expressed as median (interquartile range [IQR]) and categorical variables will be expressed as a number
- 95% confidence intervals will be calculated for the primary outcome
- Group comparisons will be analyzed by the Wilcoxon rank sum test or  $\chi^2$  test
- The placebo arm will be used as a reference group when calculating treatment effects
- Differences between rates of clinical improvement will be calculated using unadjusted ordinal logistic regression or Cox proportional hazard models
- Statistical analyses will be conducted using XLSTAT version 2020.5.1 (Addinsoft, Inc.)

#### **II. Statistical Hypotheses:**

The primary endpoint is the distribution of clinical assessments on the COVD-19 ordinal scale at day 14. The primary outcome will be analyzed using the Wilcoxon rank sum test.

The Null Hypothesis (H<sub>0</sub>) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 male subjects treated with Proxalutamide is equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 male subjects treated with the Proxalutamide placebo

The Alternative Hypothesis (H<sub>A</sub>) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 male subjects treated with Proxalutamide is not equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 male subjects treated with the Proxalutamide placebo

Mathematically written as:

$$H_0: P(X > Y) = P(Y > X)$$



 $H_A: P(X>Y) \neq P(Y>X)$ 

Where X and Y are randomly selected clinical assessments from the two treatment arms in the study.

#### **III. Primary Efficacy Analysis:**

- The non-parametric Wilcoxon rank sum test (Mann Whitney U) will be used to assess the primary end point.
- P-values <0.05 will be considered significant. All statistical analysis will be based on the intent-to-treat (ITT) population. All missing data will be described.

## 7.2 Sample Size Estimates

### Assumptions:

- The sample size estimation is based on the results reported in the placebo arm of the Adaptive COVID-19 Treatment Trial (NCT04280705)
- On day 15, 61% of subjects in NCT04280705 placebo group remained hospitalized.
- The odds ratio of improvement in the ordinal scale in the Proxalutamide arm compared to the Proxalutamide placebo is at least 2.0
- The study has two arms with randomization at 1:1 ratio
- 90% power to detect an odds ratio of 2.0 using a two-tailed test with a type I error rate of 5%
- According to NCT04280705 protocol "The sample size to detect a given odds ratio for 1:1 randomization using a 2-tailed test at level  $\alpha$  is estimated by the equation below.  $\lambda$  is the log odds ratio,  $p_i$  is the overall probability (combined over both arms) of being in the ith category of the K ordinal outcomes, and  $z_{\alpha/2}$  and  $z_{\beta}$  are the  $1 \alpha/2$  and  $1 \beta$  quantiles of the standard normal distribution."

$$\frac{12(z_{\alpha/2}+z_{\beta})^{2}}{\lambda^{2}(1-\sum_{i=1}^{K}p_{i}^{3})'}$$

- The estimated distribution is based on NCT04280705 protocol scenario 4
- 3.5% of the subjects will not complete the study based on NCT04280705

#### Sample Size Estimate:

Based on the assumptions above, we calculated that at a minimum we would need to recruit 294 subjects i.e., 147 subjects in each arm



## 7.3 Subject Population(s) for Analysis

- The primary analysis will be based on the intent-to-treat (ITT) population. The data from all subjects enrolled in the study will be analyzed.
- The safety analysis will be based on a modified intent-to-treat (MITT) population i.e., subjects who received at least one dosage of the interventional treatment.
- Subgroup analysis based on: 1) age stratification; and 2) androgen status as defined by the "Gabrin sign" will be conducted for the primary and secondary outcomes.

## 7.4 Interim Analysis

Interim efficacy and safety data will be made upon recruitment of 50% of the subjects.

#### 7.5 Termination Criteria

Upon occurrence of any one of the events listed below, the study will terminate or be modified accordingly:

- Completion of the study by a sufficient number of subjects (294 subjects) to reach our confidence level
- Termination of Arm 1: Serious adverse event due to treatment with Proxalutamide
- Substantial evidence of treatment difference between the arms. The study design will be modified to an open-label study.

## 7.6 Accountability Procedure

The data will be analyzed by a bio-statistics expert. The data will also be independently verified by an outside expert consultant.

## 7.7 Deviation Reporting

No deviation from the plan will be implemented without the prior review and approval of the EC/IRB.

## 8 Direct Access to Source Data/Documentation

The PI and hospital will permit trial-related monitoring, audits, IRB/IEC(s) review and regulatory inspection(s) by providing direct access to source data/documentation.

## 9 Quality Control and Quality Assurance

Every effort will be made to keep staff assignments consistent throughout the entire study. The PI who assesses the subject at baseline should follow the subject throughout the completion of the study. This will ensure that this study is conducted – and that data is generated, documented (recorded), and reported - in compliance with this protocol, with


GCP, and any other applicable regulatory requirements. The study monitor will audit the study procedures and CRFs throughout the study.

## 10 Ethical Considerations

This study will be conducted according to US and international standards of Good Clinical Practice (FDA regulations 21 CFR 312 for IND studies and FDA guidance E6) for all studies. Applicable government regulations and hospital research policies and procedures will also be followed.

This protocol and any amendments will be submitted to the Institutional Review Board (IRB) for formal approval to conduct the study. The decision of the IRB concerning the conduct of the study will be made in writing to the investigator.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB. The formal consent of a subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. This consent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

# 11 Data Handling and Record Keeping

During enrollment, each subject will be assigned a number. The numbers will be consecutive starting at 001.

During enrollment a record will be created for each subject. Each record will contain the subject's demographics, subject's efficacy parameters and any adverse events or study related information.

The subjects' records will be stored and handled in the same manner as the PI's patients' records.

The study monitor will keep a separate record at the monitor's office of each subject's identification number, the treatment administered to the subject (arm assignment), outcomes and any laboratory results.

No other data will be recorded. No personal information will be kept outside the study site.

Data compiled at the end of the study will not include any information that can be used to identify individuals.

The site will keep all subject records for a minimum of 3 years after the completion of the study.



# 12 Finance and Insurance

The Principal Investigator will be responsible for the cost of study. The site carries insurance for accidental injury. There is no other insurance.



## APPENDIX 1

# Drugs that should be used cautiously with Proxalutamide

## Strong CYP3A4 inducer

Avamibe, Carbamazepine, Phenytoin, Rifampicin, Mitotan, Nevirapine, Phenobarbital, Rifabutin, Rifapentine, St. John's wort, Alfentanil, Ryclosporin, Dihydroergotamine / Ergotamine, Fentanyl, Irinotecan, Pimozit, Quinidine, Sirolimus, Tacrolimus

#### Moderate CYP3A4 inducer

Smacet, Tavern, Bosentan, Efaviron, Etruverin, Lopinavir, Modafinil, Nafcillin, Thalidazine, Tiranavir, Ritonavir

# Strong CYP3A4 inhibitor

Posidovir, Clarithromycin, Conivatan, Indinavir, Itraconazole, Ketoconazole, lopinavir / Ritonavir, Mibedil, Nefazodone, Nefenavir, Posaconazole, Ritonavir, Saquinavir, Trapivir, Taliomycin, Voriconazole, Etigavir / Ritonavir, Fluconazole, Tiranavir / Ritonavir, Acetamycin

#### **Moderate CYP3A4 inhibitors**

Apronavir, Aripitan, Azanavir, Casopitam, Cimetidine, Ciprofloxacin, Clazotinib, Cyclosporin, Dalunavir, Diltiazem, Dronedarone, Erythromycin, Imatinib, Tofesoyang, Verapamil

#### Sensitive CYP3A4 substrates

Remifentanil, Aripiptam, Budesonide, Buspirone, Conivatan, Daphnesin, Darunavir, Dasatinib, Dronedarone, Eletroptan, Eplerenone, Everolimus, Felodipine, Indinavir, Fluticasone, Lopinavir, Lovastatin, Lulasidone, Maravelo, Midazolam, Nisoldipine, Quetiapine, Saquinavir, Sildenafil, Simvastatin, Sirolimus, Tolvaptan, Tiranavir, Triazolam, Vardenafil

## Narrow therapeutic index CYP3A4 Substrate

Astemizole, Cisapride, Cyclosporine, Dihydroergotamine, Fentanyl, Pethidine, Quinidine, Tacrolimus, Terfenadine

#### Sensitive CYP2D6 substrates






Tomoxetine, Decipamine, Dextromethorphan, Metoprolol, Nebeprolol, Perphenazine, Tolterodine, Venlafaxine, Avamibe, Carbamazepine, Phenytoin sodium, Rifampicin

# Narrow therapeutic index CYP2D6 Substrate

Thioridazine



| | Revision History | | | |
|---|---|---|---|---|
| Revision | <b>Description of Change</b> | | Date | Signature |
| 1 | New draft release | Andy Goren | Dec 27, 2020 | |
| 2 | | | | |



# CLINICAL STUDY PROTOCOL

Proxalutamide (GT0918)
Treatment for Hospitalized
COVID-19 Patients

## **Proprietary and Confidential**

The information contained in this document is confidential and proprietary to Applied Biology, Inc. It is offered with the express agreement that you will not disclose this document to any other person(s), or discuss the information contained herein or make reproduction by any means electronic or mechanical, or use it for any purpose other than the evaluation of the proposed clinical study for approval by an Institutional Review Board.



## **PROTOCOL NAME:**

Clinical Study: Proxalutamide Treatment for Hospitalized COVID-19 Patients

## PROTOCOL IDENTIFYING NUMBER:

**KP-DRUG-SARS-003** 

## **PROTOCOL VERSION NUMBER:**

8.0

#### **PROTOCOL VERSION DATE:**

February 1, 2021



#### GENERAL INFORMATION

## Name and address of the person(s) authorized to sign the protocol and amendments

Andy Goren, MD Flavio A. Cadegiani, MD, MSc, PhD Carlos Wambier, MD

### Name and address of study monitor

Carlos Wambier, MD

Name, title, address and telephone number(s) of the medical expert for the trial



# Name and title of the investigator(s) and sub-investigators responsible for the trial with address and phone number(s)

Flavio A. Cadegiani, MD, MSc, PhD Andy Goren, MD Carlos Wambier, MD

#### Principal Investigator (s)

Flavio A. Cadegiani, MD, MSc, PhD Andy Goren, MD

#### **Site Supervisor**

Andy Goren, MD

## **Investigator Assistant**

**TBD** 



# Protocol signature page Investigator's Agreement

Clinical Study: Proxalutamide Treatment for Hospitalized COVID-19 Patients

The information contained in this document is CONFIDENTIAL and, except to the extent necessary to obtain informed consent, may not be disclosed unless such disclosure is required by government regulation or state/local customs or law. Persons to whom the information is disclosed must be informed that the information is CONFIDENTIAL and not be further disclosed by them. By my signature below I agree to conduct this clinical study in accordance with the protocol, Good Clinical Practice, the Declaration of Helsinki, government regulations and state/local customs or laws, including those applying to institutional/ethics review and informed consent. I have read the protocol. I agree to ensure the confidentiality of my patients; however I agree to make available to the CROs, the Sponsor of this clinical study, relevant regulatory authorities, my patients' medical records. I am aware of my responsibilities as investigator as provided to me by the CROs.

| Name | Signature | Date |
|-----------------------------------|-----------|------|
| Flavio A. Cadegiani, MD, MSc, PhD | | |
| Daniel Fonseca, MD | | |



# **TABLE OF CONTENTS**

| 1. | BACK | GROUND | 8 |
|----|-------|-----------------------------------------------|----|
| | 1. | Overview | 8 |
| | 1.1. | Investigational Drug | 9 |
| | 1.1. | Pre-Clinical and Prior Clinical Data | 10 |
| | 1.1.1 | . Prior Pre-Clinical and Clinical Safety Data | 10 |
| | 1.2. | Risks/Benefits | 23 |
| | 1.3. | Trial Conduct | 23 |
| | 1.4. | Population | 23 |
| | 1.5. | Literature | 23 |
| 2. | TRIAL | OBJECTIVES | 25 |
| 3. | TRIAL | DESIGN | 25 |
| | 3.1 | Primary Study Endpoints/Secondary Endpoints | 25 |
| | 3.2 | Study Design/Type | 26 |
| | 3.3 | Randomization | 27 |
| | 3.4 | Records | 28 |
| | 3.5 | Duration | 28 |
| | 3.6 | Discontinuation | 28 |
| | 3.7 | Product Accountability | 28 |
| | 3.8 | Data Identification | 28 |
| 4. | SELEC | CTION AND WITHDRAWAL OF SUBJECTS | 29 |
| | 4.1 | Inclusion Criteria | 29 |
| | 4.2 | Exclusion Criteria | 29 |
| | 4.3 | Subject Withdrawal | 30 |

# CONFIDENTIAL



| | | | 6 Page |
|----|--------|---------------------------------------|----------|
| | 4.4 | Treatment of Subjects | 31 |
| | 4.5 | Medication | 31 |
| | 4.6 | Monitoring for subject compliance | 31 |
| 5 | ASSESS | SMENT OF EFFICACY | 31 |
| | 5.1 | Efficacy Parameters | 31 |
| | 5.2 | Method and Timing | 32 |
| 6 | ASSESS | SMENT OF SAFETY | 33 |
| | 6.1 | Safety Parameters | 33 |
| | 6.2 | Method and Timing | 33 |
| | 6.3 | Adverse Events | 34 |
| 7 | STATIS | STICAL PLAN | 38 |
| | 7.1 | Statistical Methods | 38 |
| | 7.2 | Sample Size Estimates | 39 |
| | 7.3 | Subject Population(s) for Analysis | 40 |
| | 7.4 | Interim Analysis | 40 |
| | 7.5 | Termination Criteria | 40 |
| | 7.6 | Accountability Procedure | 40 |
| | 7.7 | Deviation Reporting | 40 |
| 8 | DIREC | T ACCESS TO SOURCE DATA/DOCUMENTATION | 40 |
| 9 | QUALI | TY CONTROL AND QUALITY ASSURANCE | 41 |
| 10 | ETHI | CAL CONSIDERATIONS | 41 |
| 11 | DATA | HANDLING AND RECORD KEEPING | 41 |
| 12 | FINA | NCE AND INSURANCE | 42 |



#### **List of Abbreviations**

CFR Code of Federal Regulations

CRF Case Report Form

FDA Food and Drug Administration

GCP Good Clinical Practice

IRB Institutional Review Board

EC Ethics Committee

HCP Healthcare Professional

CDC US Center for Disease Control

SAE Serious Adverse Event

AE Adverse Event

ARDS Acute Respiratory Distress Syndrome

UP Unanticipated Problem



# 1. Background

#### 1. Overview

During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%). Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2).<sup>3–5</sup> TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro.<sup>6</sup> Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.<sup>7</sup>

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene.<sup>8-10</sup> In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor.<sup>10</sup> Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males.<sup>11</sup>

Previously, we have reported the results from two retrospective cohort analysis demonstrating the protective effect of 5-alpha-reductase inhibitors (5ARi) for men with COVID-19.<sup>17</sup> In a study of 77 men hospitalized with COVID-19 we found among men taking 5ARis, 8% were admitted to the ICU compared to 58% of men not taking 5ARis (P = 0.0015). In the cohort, 5ARis were associated with reduced risk for ICU admissions RR 0.14 (95% CI: 0.02–0.94).<sup>17</sup> Similarly, we have demonstrated that the frequency of COVID-19 symptoms was drastically reduced for men using 5ARis in an outpatient setting. A statistically significant (p<0.05) reduction in the frequency of 20 of the 29 clinical symptoms was observed in AGA men using 5ARis compared to AGA men not using 5ARis. For example, 38% and 2% of men presented with low-grade fever, 60% and 6% with dry cough, and 88% and 15% reported anosmia in the non-5ARi and 5ARi groups, respectively.<sup>18</sup>

One limitation of 5ARis is the time course required to achieve systemic DHT reductions. As such, we explored the use of a novel second generation androgen receptor antagonist Proxalutamide as a means for rapid reduction in AR activity. Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as



exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide. Because of the dual mechanism of action, it is expected to be a more effective and less toxic second-generation anti-androgen drug therapy. Clinical evidence has demonstrated that Proxalutamide lowers AR expression and activity. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells. In addition, none of the 5ARis currently approved by the US FDA have been tested in phase I studies. As such, thet are not recommended for women. Phase I studies for Proxalutamide have been successfully completed in men and women.

In December 2020, we completed a double-blinded, randomized, prospective, investigational study of Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429). The length of the study was 30 days. Proxalutamide was administered 200mg q.d. for 15 days. Men enrolled in the study were 50 years and older. Two hundred and sixty two men completed the study. 134 men were assigned to the Proxalutamide group and 128 men were assigned to the control group. Thirty five subjects were hospitalized in the control group compared to zero in the Proxalutamide group. The proportion of COVID-19 patients hospitalized was significantly different between the Proxalutamide and control arms;  $\chi^2(1) = 42.051$ , p<.0001. The difference in proportions was 27.30% with a 95%CI: [19.79%, 35.59%]. No subject receiving Proxalutamide died compared to 2 (1.56%) in the control group. There were no treatment related adverse event reported during the course of the study.

Based on the results of the Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients study (NCT04446429), the purpose of this study is to assess the efficacy and safety of Proxalutamide as a treatment for hospitalized COVID-19 male and female patients.

# 1.1. Investigational Drug

#### Proxalutamide (300 mg) q.d.

| Chemical Name | 4-[4,4-dimethyl-3-[6-[3-(2-oxazolyl)propyl]-3-pyridinyl]-5-oxo-2-thioxo-1-imidazolidinyl]-3-fluoro-2-(trifluoromethyl)-benzonitrile |
|---|---|
| CAS Registry No. | 1398046-21-3 |
| Company Code | GT0918 |
| Chemical Structure | N S N N N N N N N N N N N N N N N N N N |
| Molecular Formula | $C_{24}H_{19}F_4N_5O_2S$ |
| Relative Molecular Mass | 517.50 |



Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide. Because of the dual mechanism of action, it is expected to be a more effective and less toxic second-generation anti-androgen drug therapy. Clinical evidence has demonstrated that Proxalutamide lowers AR expression and activity. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells.

The Proxalutamide tablets (100mg per tablet) will be manufactured by:

TOT BIOPHARM International Company Limited. No. 120 changyang Street, Suzhou Industrial Park, Suzhou City, Jiangsu Province, China

#### 1.1. Pre-Clinical and Prior Clinical Data

#### 1.1.1. Prior Pre-Clinical and Clinical Safety Data

No prior pre-clinical safety data exists as to the use of Proxalutamide for the treatment of COVID-19; however, pre-clinical studies have been conducted in support of the US FDA IND approval of Phase-1 human trials of Proxalutamide in castration resistant prostate cancer and metastatic breast cancer. Selected pre-clinical animal studies conducted with Proxalutamide are provided below.

#### Tissue Distribution and Excretion of GT0918 in Rats

The tissue distribution of GT9018 in male SD rats was determined at 0.5, 3 and 12 hours following an oral single administration (20 mg/kg). Proxalutamide was extensively distributed to most of the tissues/organs with high concentrations found in fat tissue and liver, followed by stomach, pancreas and intestine in rats. Proxalutamide distribution was also observed in bone marrow in rats. Peak Proxalutamide concentrations were achieved in most tissues at 3 hours following the administration and a certain degree of elimination was observed in these tissues at 12 hours following the administration.

The excretion profiles (bile, urine and feces) following a single oral dose of Proxalutamide (20 mg/kg) to 6 male SD rats was studied. The data indicated that following a single oral administration of Proxalutamide to rats, the cumulative fractional excretion of Proxalutamide in bile within 36 hours was  $0.010 \pm 0.006\%$ , the cumulative

fractional excretion of Proxalutamide in urine within 72 hours was  $0.014 \pm 0.009\%$  and the cumulative fractional excretion of Proxalutamide in feces within 72 hours was  $10.785 \pm 4.547\%$ . Proxalutamide was mainly excreted in the feces (about 10%) and in trace amounts through bile and urine (0 to 0.1%) in rats.



#### Pharmacokinetic Profiles of Proxalutamide in SD Rats

Pharmacokinetic properties of Proxalutamide were studied in SD rats following single oral dosing at 10, 20, 40 and 80 mg/kg, single IV dosing at 5 mg/kg and repeated PO dosing at 20 mg/kg daily for 8 consecutive days. After single oral dosing, Proxalutamide reached maximal plasma concentrations in 3 to 5 hours and then decreased with the elimination half-life 2.0 to 2.5 hours. Both AUC and Cmax were proportional to dose. The absolute bioavailability was 74 - 100%. After repeated dosing for 8 days, AUC and Cmax increased about 50% comparing to single dose at the same level, indicating some drug accumulation after repeated dosing.

## Pharmacokinetic Profiles of Proxalutamide in Beagle Dogs

Pharmacokinetic properties of Proxalutamide were studied in Beagle dogs following single oral dosing at 2, 5 and 10 mg/kg under fasting conditions, single IV dosing at 1 mg/kg, a single oral dosing at 20 mg/kg (with two different API processes) under fed conditions, and repeated PO dosing at 20 mg/kg daily for 7 consecutive days. After single oral dosing, Proxalutamide reached maximal plasma concentrations in 2 to 2.5 hours and then decreased with the elimination half-life 9.5 to 11.8 hours. Both AUC and Cmax were proportional to dose. The absolute bioavailability was 36.5 – 52.5%. Under fed conditions, Cmax markedly decreased about 60% with Tmax increase from 3 hours to 8.3 hours but slightly increased in AUC compared to those respective PK parameters under fasting conditions at the same dose. After repeated dosing for 8 days, AUC and Cmax increased about 70% and 150%, respectively comparing to single dose at the same level, indicating drug accumulation after repeated dosing.

#### 1.1.2 Prior Clinical Safety Data

# <u>Study 1: Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429)</u>

A double-blinded, randomized, prospective, investigational study of Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429) was completed in December 2020. The length of the study was 30 days. Proxalutamide was administered 200mg q.d. for 15 days. Men enrolled in the study were 50 years and older. Two hundred and sixty two men completed the study. 134 men were assigned to the Proxalutamide group and 128 men were assigned to the control group. Thirty five subjects were hospitalized in the control group compared to zero in the Proxalutamide group. The proportion of COVID-19 patients hospitalized was significantly different between the Proxalutamide and control arms;  $\chi 2$  (1) = 42.051, p<.0001. The difference in proportions was 27.30% with a 95%CI: [19.79%, 35.59%]. No subject receiving Proxalutamide died compared to 2 (1.56%) in the control group. There were no treatment related adverse event reported during the course of the study.



#### Study 2: Phase 1 study in 16 males with prostate cancer.

The data from the study was published in a peer review journal. The identifier GT0918 was used to denote Proxalutamide. The abstract from the publication is below:

Abstract Purpose: We conducted preclinical experiments and phase I clinical trial to investigate the safety, pharmacokinetics (PK) and antitumour effects of GT0918 in castration- resistant prostate cancer (CRPC).

Experimental design: An androgen receptor (AR) competitive binding assay was performed, followed by evaluation of GT0918 on AR protein expression. The efficacy of GT0918 was investigated in a castration-resistant xenograft model. A phase I dose-escalation study of GT0918 in CRPC was also carried out to evaluate its safety, PK and antitumour efficacy. Results: GT0918 was demonstrated to inhibit the binding of androgen to AR more potently than MDV3100, and to effectively reduce the AR protein level. GT0918 inhibited the tran-scriptional activity of wild-type AR and AR with clinically relevant ligand-binding domain mutations. Furthermore, GT0918 significantly inhibited the growth of prostate cancer. A total of 16 patients was treated with GT0918 at five dose levels. Among these 16 patients, 10 and 2 patients, respectively, completed a three-cycle and sixcycle treatment, in which MTD was not reached. All the treatment-related adverse events were grade I, including hypercholesterolemia, hypertriglyceridemia, fatigue and anemia. PK parameters showed that drug exposure increased with dose proportionally from 50 to 300 mg and a saturation was observed between 300mg and 400 mg.

The most significant adverse events from the study are summarized in the following table:

| Table 2 | | | |
|---|---|---|---|
| Most common adverse | events of GT0918 by | dose (multiple-dose | period, ≥2 cycles). |

| Adverse event | 50 mg (n=2) | | 100 mg (n = 4) | | 200 mg (n = 3) | 3) | 300 mg (n = 1) | 3) | 400 mg (n = 400 mg) | Total $(n = 16)$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Drug-<br>related | Drug-<br>irrelative | Drug-<br>related | Drug-<br>irrelative | Drug-related | Drug-<br>irrelative | Drug-related | Drug-irrelative | Drug-related | Drug-<br>irrelative | Drug-<br>related | Drug-<br>irrelative |
| Blood and lymphatic diseases | | | | | | | | | | | | |
| Anaemia | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 |
| Heart diseases | | | | | | | | | | | | |
| Coronary artery disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Visual diseases | | | | | | | | | | | | |
| Eve discomfort | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Gastrointestinal diseases | | | | | | | | | | | | |
| Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |
| Systemic diseases | | | | | | | | | | | | |
| Chest pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| Peripheral oedema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 |
| Abnormal examination results | | | | | | | | | | | | |
| Prolonged coagulation indicators | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| OT interval extension | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| LDH increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| ALP increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |
| Metabolic and nutritional diseases | | | | | | | | | | | | |
| Hypercholesterolemia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 |
| Malnutrition | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Musculoskeletal and connective tissue diseases | | | | | | | | | | | | |
| Arthralgia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Neurological diseases | | | | | | | | | | | | |
| Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 |
| Urinary diseases | | | | | | | | | | | | |
| Haematuria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| Vascular diseases | | | | | | | | | | | | |
| Aortic aneurysm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
| Hot flushes | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |

LDH, lactate dehydrogenase; ALP, alkaline phosphatase.

Table 2



## Study 3: Phase 1 study conducted in 40 males with prostate cancer.

A summary of the study is provided below:

Demographics: All 40 patients in the Safety Analysis Set were male with the mean age at 70.1 years. Three (7.5%) patients were Hispanic or Latino and 37 (92.5%) were not Hispanic or Latino. Thirty-five (87.5%) patients were white, 4 (10%) were black or African American and 1 (2.5%) was Asian. Of the 40 patients with mCRPC tumors, all patients (100%) had received at least two lines of hormone therapies, with 11 (27.5%) having 3 lines and 20 (50%) having 4 lines or more. Most patients (70%) had also undergone chemotherapies, with 20 (50%) receiving one line and 8 (20%) receiving 2 or more lines of chemotherapies.

Disposition: The distribution of 40 patients by dose cohort was as follows: 3 at the 50 mg, 6 at the 100 mg, 6 at the 200 mg, 7 at the 300 mg, 7 at the 400 mg, 6 at the 500 mg and 5 at the 600 mg per day dose levels. Of the 40 patients, 1 (2.5%) did not complete 1 cycle, 14 (35%) completed 1 cycle, 10 (25%) completed 2 cycles, 3 (7.5%) completed 3 cycles, 3 (7.5%) completed 4 cycles, 5 (12.5%) completed 5 cycles, and 4 (10%) completed at least 6 cycles of treatment. The primary reason for discontinuation was progressive disease (28/40 patients, 70%). Other discontinuation reasons included the following: unacceptable toxicity or AE (6/40, 15%), withdrawal of consent (4/40, 10%) and patient lost to follow-up (2/40, 5%).

Efficacy: Of the 40 patients, no PSA response with more than 50% reduction from baseline was observed. CR or PR are not required as per phase 1 study data analyses. Treating physicians will do imaging scan to see if patients have with SD allowing for continuing the treatment. The mean number of dosing duration was 12.5 weeks (87.6 days) across all dose cohorts from 50 mg/day to 600 mg/day, and the mean dosing duration for individual dose cohorts ranged from 8.3 weeks (57.7 days) to 15.6 weeks (109.4 days). Patients with treatment duration longer than 22.9 weeks (160 days) were from the following dose cohorts: 1 in the 50 mg/day, 1 in the 100 mg/day, and 2 in the 400 mg/day cohorts. A total of 9 patients had completed between 4 and 6 cycles (28 days per cycle) of treatment, belonging to these dose cohorts: 200 mg/day (1/6), 400 mg/day (4/7), 500 mg/day (2/6), and 600 mg/day (2/5).

Safety: The results from this study showed that the safety profile of GT0918 was generally favorable in patients with mCRPC whose disease progressed after multi-lines of therapies. The mean number of dosing duration was 87.6 days across all dose cohorts from 50 mg/day to 600 mg/day, and the mean dosing duration for individual dose cohorts ranged from 57.7 to 109.4 days. Of the 40 patients, 39 (98%) experienced at least 1 TEAE during the study, with the most frequent AEs being fatigue, nausea, decreased appetite, anemia, weight decrease, diarrhea, constipation, back pain and dizziness. Most of patients reported TEAEs that were considered related to the study drug, with the most common drug-related AEs being fatigue (42.5%), decreased appetite (20%), nausea (15%), dizziness (12.5%), constipation (12.5%), anemia (10%), weight decrease (10%), dysgeusia (10%), and diarrhea (7.5%). Most TEAEs were Grade 1 or 2. Twenty patients across all dose cohorts reported TEAEs of Grade 3 or higher. Each individual TEAE of Grade 3 or higher occurred sporadically in 1 or 2 patients, except for the following: anemia (7/40), fatigue (5/40) and sepsis (3/40). The majority of Grade 3 or higher TEAEs were considered not related to the study drug. Overall, nine patients (9/40, 22.5%)



reported at least one SAE. The nine patients were distributed in nearly all dose cohorts except the 100 mg/day cohort. The majority of SAEs were Grade 3 or 4, and two Grade 5 deaths were reported. Both deaths were due to disease progression and they were not related to the study drug. Most SAEs were not drug-related, except for one event of Grade 4 increased creatine phosphokinase (CK). Five patients with SAEs, including sepsis, worsening dehydration, pneumonia and increased CK, were permanently discontinued from the study. Other drug-related AEs that led to study discontinuation included: fatigue (Grade 3 and Grade 2), anemia (Grade 3) and decreased white blood cell (Grade 3). No DLT was reported in any of the dose cohort. Therefore, MTD was not established in this study. Overall, GT0918 was generally well-tolerated in mCRPC patients.

A summary of AEs are given in the following tables:

Table 12.3 Overview of Treatment-Emergent Adverse Events, Safety Analysis Set

| | | | | Esc | al | ation Coh | OI | t | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 50 mg/<br>(N=:<br>n (S | 1) | (N=6)<br>n (%) | 200 mg/day<br>(N=6)<br>n (%) | 30 | 0 mg/day<br>(N=7)<br>n (%) | 40 | 00 mg/day<br>(N=7)<br>n (%) | 50 | 0 mg/day<br>(N=6)<br>n (%) | 60 | 0 mg/day<br>(N=5)<br>n (%) | | Total<br>(N=40)<br>n (%) |
| Adverse Events | 3 (100 | .0%) | 5 (83.3%) | 6 (100.0%) | 7 | (100.0%) | 7 | (100.0%) | 6 | (100.0%) | 5 | (100.0%) | 39 | (97.5% |
| Drug-Related Adverse Events | 0 | | 3 (50.0%) | 4 (66.7%) | 6 | (85.7%) | 6 | (85.7%) | 6 | (100.0%) | 5 | (100.0%) | 30 | (75.0% |
| Deaths | 0 | | 0 | 0 | 1 | (14.3%) | 1 | (14.3%) | | 0 | | 0 | 2 | (5.0%) |
| Serious Adverse Events | 1 (33 | 3%) | 0 | 1 (16.7%) | 2 | (28.6%) | 3 | (42.9%) | 1 | (16.7%) | 1 | (20.0%) | 9 | (22.5%) |
| Drug-Related Serious Adverse<br>Events | 0 | | 0 | 0 | | 0 | | 0 | 1 | (16.7%) | | 0 | 1 | (2.5%) |
| Adverse Events Leading to<br>Permanent Discontinuation of<br>Study Drug | 0 | | 0 | 0 | 3 | (42.9%) | 2 | (28.6%) | 2 | (33.3%) | 2 | (40.0%) | 9 | (22.5%) |
| Drug-Related Adverse Events<br>Leading to Permanent<br>Discontinuation of Study Drug | 0 | | 0 | 0 | 2 | (28.6%) | | 0 | 2 | (33.3%) | 2 | (40.0%) | 6 | (15.0%) |
| Grade 3 or Higher Treatment-<br>Emergent Adverse Events | 2 (66 | 7%) | 1 (16.7%) | 3 (50.0%) | 3 | (42.9%) | 7 | (100.0%) | 2 | (33.3%) | 2 | (40.0%) | 20 | (50.0% |



Table 12.4 Treatment-Emergent Adverse Events by System Organ Class >20%, Safety Analysis Set

| | | | | | | Esc | al | ation Col | oz | t | | | | | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | | GT0918<br>0 mg/day<br>(N=3)<br>n (%) | | GT0918<br>0 mg/day<br>(N=6)<br>n (%) | 20 | GT0918<br>00 mg/day<br>(N=6)<br>n (%) | 30 | GT0918<br>00 mg/day<br>(N=7)<br>n (%) | 40 | GT0918<br>00 mg/day<br>(N=7)<br>n (%) | 50 | GT0918<br>00 mg/day<br>(N=6)<br>n (%) | | GT0918<br>00 mg/day<br>(N=5)<br>n (%) | | Total<br>(N=40)<br>n (%) |
| Overall | 3 | (100.0%) | 5 | (83.3%) | 6 | (100.0%) | 7 | (100.0%) | 7 | (100.0%) | 6 | (100.0%) | 5 | (100.0%) | 39 | (97.5% |
| General Disorders And<br>Administration Site Conditions | 2 | (66.7%) | 3 | (50.0%) | 4 | (66.7%) | 6 | (85.7%) | 3 | (42.9%) | 6 | (100.0%) | 4 | (80.0%) | 28 | (70.0% |
| Fatigue | 2 | (66.7%) | 1 | (16.7%) | 2 | (33.3%) | 4 | (57.1%) | 3 | (42.9%) | 6 | (100.0%) | 3 | (60.0%) | 21 | (52.5% |
| Musculoskeletal And Connective | 2 | (66.7%) | 3 | (50.0%) | 4 | (66.7%) | 5 | (71.4%) | 7 | (100.0%) | 4 | (66.7%) | 1 | (20.0%) | 26 | (65.0% |
| Arthralgia<br>Back Pain | 1 | (33.3%) | 2 | 0<br>(33.3%) | 3 | (50.0%) | | (14.3%)<br>(57.1%) | | (28.6%)<br>(28.6%) | 2 | 0<br>(33.3%) | | 0 | | (17.5%)<br>(25.0%) |
| Gastrointestinal Disorders | 1 | (33.3%) | 3 | (50.0%) | 4 | (66.7%) | 3 | (42.9%) | 5 | (71.4%) | 5 | (83.3%) | 4 | (80.0%) | 25 | (62.5% |
| Constipation<br>Diarrhoea | | 0 | 2 | (33.3%) | | (33.3%)<br>(16.7%) | | | | (28.6%)<br>(71.4%) | | | | 0 | | (25.0%) |
| Nausea | 1 | (33.3%) | 1 | (16.7%) | 2 | (33.3%) | 1 | (14.3%) | 4 | (57.1%) | 2 | (33.3%) | 2 | (40.0%) | 13 | (32.5% |
| Nervous System Disorders | 2 | (66.7%) | | | 4 | (66.7%) | | A STATE OF THE PARTY OF THE PAR | | | | (33.3%) | | | | |
| Dizziness | | U | 1 | (16.7%) | | U | - | (20.04) | ٥ | (12.98) | - | (33.3%) | 1 | (20.04) | 9 | (22.5%) |

Table 12.4 Treatment-emergent Adverse Events by System Organ Class >20%

page 2 of 2

| Escalation Cohort | | | | | | | | Total |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | GT0918<br>50 mg/day<br>(N=3)<br>n (%) | GT0918<br>100 mg/day<br>(N=6)<br>n (%) | GT0918<br>200 mg/day<br>(N=6)<br>n (%) | GT0918<br>300 mg/day<br>(N=7)<br>n (%) | GT0918<br>400 mg/day<br>(N=7)<br>n (%) | GT0918<br>500 mg/day<br>(N=6)<br>n (%) | GT0918<br>600 mg/day<br>(N=5)<br>n (%) | Total<br>(N=40)<br>n (%) |
| Metabolism And Nutrition<br>Disorders | 1 (33.3%) | 2 (33.3%) | 2 (33.3%) | 4 (57.1%) | 5 (71.4%) | 4 (66.7%) | 3 (60.0%) | 21 (52.5%) |
| Decreased Appetite | 0 | 1 (16.7%) | 1 (16.7%) | 2 (28.6%) | 3 (42.9%) | 3 (50.0%) | 2 (40.0%) | 12 (30.0%) |
| Investigations | 1 (33.3%) | 1 (16.7%) | 1 (16.7%) | 4 (57.1%) | 3 (42.9%) | 4 (66.7%) | 1 (20.0%) | 15 (37.5%) |
| Weight Decreased | 1 (33.3%) | 0 | 1 (16.7%) | 1 (14.3%) | 3 (42.9%) | 3 (50.0%) | 1 (20.0%) | 10 (25.0%) |
| Respiratory, Thoracic And<br>Mediastinal Disorders | 2 (66.7%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 4 (57.1%) | 1 (16.7%) | 2 (40.0%) | 15 (37.5%) |
| Blood And Lymphatic System<br>Disorders | 1 (33.3%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 4 (57.1%) | 1 (16.7%) | 1 (20.0%) | 13 (32.5%) |
| Anaemia | 1 (33.3%) | 1 (16.7%) | 2 (33.3%) | 3 (42.9%) | 3 (42.9%) | 1 (16.7%) | 0 | 11 (27.5%) |
| Infections And Infestations | 2 (66.7%) | 0 | 0 | 2 (28.6%) | 4 (57.1%) | 0 | 3 (60.0%) | 11 (27.5%) |
| Vascular Disorders | 0 | 3 (50.0%) | 1 (16.7%) | 2 (28.6%) | 4 (57.1%) | 0 | 1 (20.0%) | 11 (27.5%) |
| Renal And Urinary Disorders | 1 (33.3%) | 0 | 2 (33.3%) | 3 (42.9%) | 1 (14.3%) | 1 (16.7%) | 0 | 8 (20.0%) |
| Cardiac Disorders | 1 (33.3%) | 0 | 0 | 2 (28.6%) | 3 (42.9%) | 1 (16.7%) | 1 (20.0%) | 8 (20.0%) |

Study 4: Phase II dose escalating study of Proxalutamide (100-300 mg) in 108 patients with prostate cancer.

A table of adverse events observed in the trial are described below.


This material is the property of the Applied Biology Inc. Do not disclose or use except as authorized.

AVIA MEV



| PT name | 100 mg<br>(N=37)% | 200 mg<br>(N=35)% | 300 mg<br>(N=36)% | Total<br>(N=108)% | P |
|---|---|---|---|---|---|
| Asthenia/ fatigue | 2 (5.4) | 7 (20.0) | 14 (38.9 | 23 (21.3) | < 0.05 |
| Aspartate aminotransferase | 5 (13.5) | 5 (14.3) | 6 (16.7) | 16 (14.8) | >0.05 |
| Anaemia | 3 (8.1) | 7 (20.0) | 6 (16.7) | 16 (14.8) | >0.05 |
| Alanine aminotransferase increased | 6 (16.2) | 4 (11.4) | 4 (11.1) | 14 (13.0) | >0.05 |
| Decreased appetite | 3 (8.1) | 3 (8.6) | 8 (22.2) | 14 (13.0) | >0.05 |
| White blood cell count decreased | 2 (5.4) | 5 (14.3) | 6 (16.7) | 13 (12.0) | >0.05 |
| Proteinuria | 4 (10.8) | 4 (11.4) | 5 (13.9) | 13 (12.0) | >0.05 |
| Constipation | 1 (2.7) | 3 (8.6) | 6 (16.7) | 10 (9.3) | >0.05 |
| Oedema peripheral | 1 (2.7) | 4 (11.4) | 3 (8.3) | 8 (7.4) | >0.05 |
| Blood fibrinogen increased | 2 (5.4) | 2 (5.7) | 3 (8.3) | 7 (6.5) | >0.05 |
| Blood triglycerides increased | 5 (13.5) | 2 (5.7) | 0 | 7 (6.5) | >0.05 |
| Neutrophil count decreased | 0 | 4 (11.4) | 3 (8.3) | 7 (6.5) | >0.05 |
| Weight decreased | 1 (2.7) | 2 (5.7) | 4 (11.1) | 7 (6.5) | >0.05 |
| Hypertriglyceridaemia | 1 (2.7) | 3 (8.6) | 3 (8.3) | 7 (6.5) | >0.05 |
| Nausea | 1 (2.7) | 0 | 6 (16.7) | 7 (6.5) | < 0.05 |
| Supraventricular extrasystoles | 1 (2.7) | 3 (8.6) | 2 (5.6) | 6 (5.6) | >0.05 |
| Haematuria | 2 (5.4) | 3 (8.6) | 1 (2.8) | 6 (5.6) | >0.05 |
| Platelet count decreased | 2 (5.4) | 1 (2.9) | 2 (5.6) | 5 (4.6) | >0.05 |

Study 5: Phase I dose escalating study of Proxalutamide (100-500 mg) in 67 female patients with metastatic breast cancer positive for androgen receptor (AR+)

Background: Androgen receptor (AR) blocker has become an increased interest in the treatment of BC, in which about 60-80% patients showed AR positive. However, currently no AR blocker has been approved in mBC. GT0918 is a new chemical entity of AR blocker with possible AR down-regulation. This study is an open-label, single-center, dose escalation phase I trial to assess GT0918 in mBC female patients who have progressed after systemic treatments in China. The primary objectives are to identify the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs). The secondary objectives are to assess pharmacokinetics and pharmacodynamics of GT0918 with single and multiple dosage applications. (CTR20170757) Methods: Patients (pts) with historically confirmed mBC who had progressed after either chemotherapy, hormonal or targeted therapy, or could not tolerate currently standard therapies were eligible. With the starting dose at 100 mg of GT0918, the decision of dose escalation in the 3+3 design was based on the safety and tolerability assessments. GT0918 was administered orally once, followed by a 7-day off-treatment period for single dose PK analysis of drug elimination. Then GT0918 oral administration was resumed once daily for 28 consecutive days and multiple dose PK analysis was assessed at the end of first cycle (28 days). The first 28days on treatment (cycle 1) was defined as DLT period. Pts manifesting an objective response or stable disease and likely to have clinical benefit from continued treatment were continued on GT0918 thereafter until they experienced one of following events of intolerable toxicities, disease progression or withdrew consent. Results: 18 pts were




enrolled and treated with GT0918 since 9/6/2017 as defined in protocol at five dose levels: 100 mg (n = 3), 200 mg (n = 4), 300 mg (n = 4), 400 mg (n = 4) and 500 mg (n = 3) (as to 7/2/2019). All pts progressed more than two lines of therapies with 83.3%(15/18) pts were treated  $\geq 3$ rd lines. Out of 6 confirmed AR positive pts, two (33.3%) at 300 mg cohort had finished 17 and 19 cycles individually and continue treatment (as 7/2/19). No DLT was observed and MTD has not been reached. GT0918 related adverse events (AEs) were grade 1 or 2 as per CTCAE v4.03, including fatigue, hypertriglyceridemia, anemia, hypercholesterolemia, increased LDL, nausea, loss of appetite, increased ALT, increase of weight loss, constipation and thrombocytopenia. PK profile analysis showed that in the single-dose study, GT0918 showed a fast absorption profile. In the multiple-dose study, the steady-state serum concentration level of GT0918 and its main metabolite were attained at 21 days. Conclusions: Proxalutamide (GT0918) administrated orally once a day is well tolerated in late-stage pts. No DLT has occurred at maximum dose 500 mg. Pts with AR positive biomarker could have better clinical outcomes with GT0918 treatment. GT0918 and its main metabolite exhibited a nonlinear pharmacokinetic profile over the dose range from 100mg to 500 mg. An expanded/phase Ib in AR positive mBC pts has launched in China to evaluate the anti-tumor activity and safety of GT0918. 200 mg and 300 mg were selected for dose expansion.

#### **Drug Interactions**

Inhibition Potential Assessment of Proxalutamide on Cytochrome P450 Enzymes in Pooled Human Liver Microsomes

The inhibition of human liver CYPs: CYP1A2, CYP2C9, CYP2C19, CYP2D6, CYP2E1 and CYP3A4/5, was assessed with Proxalutamide at concentrations of 0.2, 0.8, 2, 10, 50, 100 and 200 µM. The metabolite formation from CYP catalyzed probe substrate metabolism was analyzed with LC-MS/MS. The results showed that Proxalutamide showed no significant inhibition on CYP1A2 and CYP2E1, weak inhibition on CYP2D6, CYP2C9, CYP2C19 and CYP3A (midazolam), but marked inhibition on CYP3A4 (testosterone).

The results indicate that there is an inhibitory effect of Proxalutamide on CYP3A4 in vitro and the corresponding in vivo drug interaction potential needs to be further investigated.

\*No interaction has been reported between Proxalutamide, nitazoxanide, and azithromycin.



| <b>Table 1.2.3:</b> | Inhibitory Ef | Inhibitory Effect of Proxalutamide on CYP450 Enzymes | | |
|---|---|---|---|---|
| CYP450s | Probe substrate | Characterized Metabolite | IC <sub>50</sub> ( <u>M</u> ) | |
| CYP1A2 | Phenacetin | Deethylation | Acetaminophen | >200 |
| CYP2C9 | Tolbutamide | Hydroxylation | 4-Hydroxy-Tolbutamide | 8 |
| CYP2C19 | Omeprazole | Hydroxylation | 5-Hydroxy- Omeprazole | 8 |
| CYP2D6 | Dextromethorphan | Demethylation | Dextrorphan | 5 |
| CYP3A4 | Midazolam | Hydroxylation | 1-Hydroxy-Midazolam | 56 |
| CYP3A4 | Testosterone | Hydroxylation | 6β-Testosterone | 1 |
| CYP2E1 | Chlorzoxazone | Hydroxylation | 6-Hydroxy-Chlorzoxazone | >200 |

<u>Evaluation of Cytochrome P450 Induction Potential of Proxalutamide in Human Hepatocytes</u>

Proxalutamide was evaluated for induction of drug metabolizing enzymes in primary human hepatocytes. No inductive effects on CYP1A2 and CYP3A4 were observed in the level of enzymatic activity.

Table 10: Effect of Proxalutamide on the Enzyme Activity of CYP1A2

| | Activity | of CYP1A | 2 (%) | Mean | SD | Activity compared to positive control (%) |
|---|---|---|---|---|---|---|
| Negative control | 109 | 82.4 | 108 | 100 | 15.2 | NA |
| Positive control | 1174 | 1246 | 1207 | 1209 | 36.3 | 100 |
| Proxalutamide 1 µM | 98.9 | 98.2 | 95.6 | 97.6 | 1.74 | <40 |
| Proxalutamide 10 µM | 92.3 | 98.9 | 99.6 | 96.9 | 4.01 | <40 |

| Table 11: Effect of PROXALUTAMIDE on the Enzyme Activity of CYP3A4 | | | | | | |
|---|---|---|---|---|---|---|
| Control | Activit | y of CYP3A | 4(%) | Mean | SD | Activity compared to positive control (%) |
| Negative control | 97.3 | 103 | 99.6 | 100 | 2.97 | NA |
| Positive control | 805 | 976 | 825 | 869 | 93.4 | 100 |
| Proxalutamide 1 µM | 24.2 | 26.0 | 27.7 | 26.0 | 1.73 | <40 |
| Proxalutamide 10µM | 19.7 | 21.3 | 19.4 | 20.2 | 1.05 | <40 |



## Specific Populations

### <u>Pediatric</u>

Proxalutamide pharmacokinetics have not been investigated in subjects younger than 18 years.

#### Geriatric

No dose adjustment is necessary in the elderly. The pharmacokinetics and pharmacodynamics of Proxalutamide were evaluated in 40 patients with an average age of 70.1 (Study 2, Section 1.1.2.4.).

#### Gender

Proxalutamide is not indicated for use in women. The palnned interventional study will be conducted in men only.

#### Race

The effect of race on Proxalutamide pharmacokinetics has not been studied.

#### Renal Impairment

The effect of renal impairment on Proxalutamide pharmacokinetics has not been studied.

### Hepatic Impairment

The effect of hepatic impairment on Proxalutamide pharmacokinetics has not been studied.

#### 1.1.3 Prior Pre-clinical Efficacy Data

No prior pre-clinical data exists as to the use of Proxalutamide as a treatment for COVID-19.; however, two studies highlight the possible benefit of the dual anti-androgen activity of Proxalutamide.

#### Proxalutamide inhibition of androgen binding to AR and AR protein expression

A study by Zhou et al<sup>19</sup> reported that: "GT0918 inhibited the binding of androgen to AR in a dose-dependent manner, and the Ki value of GT0918 (1.4 x 10<sup>-8</sup> M) in binding to AR was 3.4-fold lower than that of MDV3100 (4.8 x 10<sup>-8</sup> M) (Fig. 1A). It indicated that GT0918 was more potent than MDV3100 in inhibiting the binding of androgen to AR." Additionally, in cultures of C4-2B cells, "the protein expression of AR was significantly reduced by GT0918". Data depicting the inhibition androgen binding to AR and the reduced AR protein expression in C4-2B cells is shown below:





Fig. 1. GT0918 effectively decreases androgen binding to AR. (A) IC<sub>50</sub> values for GT0918 and MDV3100 in inhibiting androgen from binding to AR. (B) GT0918 reduces the protein expression of AR in C4-2B cells.

### Proxalutamide suppression ACE2 and TMPRSS2 in A549 lung cells

A study by Wu et al <sup>20</sup> reported that "In LNCaP and A549 cells, we showed that androgen induced the ACE2 and TMPRSS2 expression, and GT0918 could suppress the ACE2 and TMPRSS2 expression". The data from the study is depicted in the figure below.





#### 1.1.4 Prior Clinical Efficacy Data

# Study 1: Proxalutamide Treatment for Non-Hospitalized COVID-19 Male Patients (NCT04446429)

Proxalutimede has been studied in a prospective clinical trial as a treatment for non-hospitalized COVID-19 male patients. A summary of the study and the results are as follows:

Objective: To determine if the anti-androgen Proxalutamide is an effective treatment for men not-hospitalized due to COVID-19 disease (based on assessment of the clinical status on an 8 point ordinal scale: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities) Design: A double-blinded, randomized, prospective, investigational study of Proxalutamide as a treatment for non-hospitalized COVID-19 male patients (inclusion ordinal scale <3).

**Setting:** Outpatient centers (Brasilia, Brazil) from October 21 to December 24, 2020. Participants: Men not hospitalized due to COVID-19 disease (inclusion ordinal scale <3) **Interventions:** Proxalutamide 200mg/day, or standard of care for 15 days.

Main Outcome and Measures: Percentage of subjects hospitalized due to COVID-19 [Time Frame: 30 days]

**Results:** A total of 268 men were included and completed the trial; 134 men were randomized to the Proxalutamide group, and 134 men were randomized to the control group. Data is summarized in Table 1.4.1. A statistically significant difference (p<0.001) in the percentage of subjects hospitalized due to COVID-19 was observed in men taking Proxalutamide compared to the standard of care. The percentage of men hospitalized were 2.2% and 26% in the Proxalutamide and control groups, respectively. No subject receiving Proxalutamide died versus 2 (1.56%) in the control group. **Conclusions and Relevance:** Non-hospitalized COVID-19 male patients (inclusion ordinal scale <3) treated with Proxalutamide, had significantly reduced rate of

Trial Registration: NCT04446429

| | Control | Proxalutamide |
|------------------|---------|---------------|
| Not Hospitalized | 99 | 131 |
| Hospitalized | 35 | 3 |
| Total | 134 | 134 |

hospitalization compared to men not receiving Proxalutamide.



Table 1.4.1 Clinical outcomes of COVID-19 male patients treated with Proxalutamide compared to standard of care.

Study 2: <u>Proxalutamide Treatment for Non-Hospitalized COVID-19 Female Patients</u> (NCT04446429)



#### 1.1.5 Justification for Dosage

According to a phase I study of Proxalutamide conducted by Zhou et al<sup>19</sup> PK parameters showed that drug exposure increased with dose proportionally from 50 to 300 mg and a saturation was observed between 300mg and 400 mg.

Further, the research team conducting the NCT04446429 study had previously administered to five COVID-19 male patients Proxalutamide at dosages as high as 400mg q.d. These patients did not qualify to be enrolled in the study due to age <50. In the assessment of the research team, these patients were at an imminent threat of hospitalization due to COVID-19. All patients have exhibited shortness of breath, coughing and oxygen saturation <=93%. A marked improvement in symptoms was observed 24 hours following administration of 400mg Proxalutamide. None of the imminent were subsequently hospitalized. No treatment related adverse events were observed.

As such, we believe that Proxalutamide 300mg q.d.is likely to provide efficacy in the treatment of hospitalized COVID-19 patients without increasing the rate of treatment related adverse events (none observed in NCT04446429)

#### 1.1.6 Other Data



The PI has not identified any additional data related to the safety or efficacy of this study.

## 1.2. Risks/Benefits

This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study to assess the efficacy of Proxalutamide as a treatment for hospitalized COVID-19 male and female patients; therefore, we assess below the risks/benefits for the proposed study.

## Benefit(s) of the Proposed Clinical Study

To-date no therapy for hospitalized COVID-19 patients has demonstrated significant clinical benefit. Proxalutamide demonstrated clinical efficacy in non-hospitalized COVID-19 patients (NCT04446429). As such, subjects enrolled in this study could potentially benefit from reduced hospitalization time as well as lower risk of experiencing progressively more severe COVID-19 related symptoms. In addition, if Proxalutamide demonstrates clinical efficacy in this study, it is likely to improve the standard of care for hospitalized COVID-19 male and female patients world-wide.

#### Risk(s) of the Proposed Clinical Study

Treatment with any drug carries risk. Treatment with Proxalutamide caries the risk of the adverse events reported in Phase I clinical trials with Proxalutamide; however, due to the short treatment duration of 14 days, we believe the risk of serious adverse events is lower than described in Phase I studies. Further, during 14 days of dosing 134 subjects with 200mg q.d. of Proxulatimde no drug related adverse events were observed.

#### 1.3. Trial Conduct

This study will be conducted in compliance with the protocol approved by the Institutional Review Board (Ethics Committee), and according to Good Clinical Practice standards. No deviation from the protocol will be implemented without the prior review and approval of the IRB (EC) except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the IRB (EC) as soon as possible.

# 1.4. Population

This is a multi-center study to be conducted at hospital sites. This exact protocol will be followed. There will be one or more PIs. The study will be approved by each hospital's Ethics Committee.

The population for this study will be hospitalized COVID-19 patients 18 years or older of any ethnicity. Approximately, 600 (300 males and 300 females) subjects who meet all the eligibility criteria will be enrolled. The estimated time from screening to end of the study for each subject is approximately 28 days.

#### 1.5. Literature

1. Guan W-J, Ni Z-Y, Hu Y, et al. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. February 2020:NEJMoa2002032. doi:10.1056/NEJMoa2002032



- 2. Goren A, Mc Coy J, Wambier CG, et al. WHAT DOES ANDROGENETIC ALOPECIA HAVE TO DO WITH COVID-19? AN INSIGHT INTO A POTENTIAL NEW THERAPY. Dermatol Ther. April 2020:e13365. doi:10.1111/dth.13365
- 3. Shieh WJ, Hsiao CH, Paddock CD, et al. Immunohistochemical, in situ hybridization, and ultrastructural localization of SARS-associated coronavirus in lung of a fatal case of severe acute respiratory syndrome in Taiwan. Hum Pathol. 2005. doi:10.1016/j.humpath.2004.11.006
- 4. Hoffmann M, Kleine-Weber H, Schroeder S, et al. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. March 2020:1-10. doi:10.1016/j.cell.2020.02.052
- 5. Glowacka I, Bertram S, Muller MA, et al. Evidence that TMPRSS2 Activates the Severe Acute Respiratory Syndrome Coronavirus Spike Protein for Membrane Fusion and Reduces Viral Control by the Humoral Immune Response. J Virol. 2011. doi:10.1128/jvi.02232-10
- 6. Heurich A, Hofmann-Winkler H, Gierer S, Liepold T, Jahn O, Pohlmann S. TMPRSS2 and ADAM17 Cleave ACE2 Differentially and Only Proteolysis by TMPRSS2 Augments Entry Driven by the Severe Acute Respiratory Syndrome Coronavirus Spike Protein. J Virol. 2014;88(2):1293-1307. doi:10.1128/JVI.02202-13
- 7. Limburg H, Harbig A, Bestle D, et al. TMPRSS2 Is the Major Activating Protease of Influenza A Virus in Primary Human Airway Cells and Influenza B Virus in Human Type II Pneumocytes. Schultz-Cherry S, ed. J Virol. 2019;93(21). doi:10.1128/JVI.00649-19
- 8. Lucas JM, Heinlein C, Kim T, et al. The Androgen-Regulated Protease TMPRSS2 Activates a Proteolytic Cascade Involving Components of the Tumor Microenvironment and Promotes Prostate Cancer Metastasis. Cancer Discov. 2014;4(11):1310-1325. doi:10.1158/2159-8290.CD-13-1010
- 9. National Institutes of Health. TMPRSS2 transmembrane serine protease 2 [ Homo sapiens (human) ] Gene ID: 7113. Gene ID: 7113, updated on 13-Mar-2020. https://www.ncbi.nlm.nih.gov/gene/7113. Published 2020. Accessed April 2, 2020. 10. Lin B, Ferguson C, White JT, et al. Prostate-localized and androgen-regulated expression of the membrane- bound serine protease TMPRSS2. Cancer Res. 1999.
- 11. Dalpiaz PLM, Lamas AZ, Caliman IF, et al. Sex Hormones Promote Opposite Effects on ACE and ACE2 Activity, Hypertrophy and Cardiac Contractility in Spontaneously Hypertensive Rats. Bader M, ed. PLoS One. 2015;10(5):e0127515. doi:10.1371/journal.pone.0127515
- 12. Gan DCC, Sinclair RD. Prevalence of male and female pattern hair loss in Maryborough. J Investig Dermatol Symp Proc. 2005;10(3):184-189. doi:10.1111/j.1087-0024.2005.10102.x 13. Goren et al. A PRELIMINARY OBSERVATION: MALE PATTERN HAIR LOSS AMONG HOSPITALIZED COVID-19 PATIENTS IN SPAIN A POTENTIAL CLUE TO THE ROLE OF ANDROGENS IN COVID-19 SEVERITY. J. Cos. Derm (accepted April 2020)
- 14. Severi G, Sinclair R, Hopper JL, English DR, McCredie MR, Boyle P, Giles GG. Androgenetic alopecia in men aged 40-69 years: prevalence and risk factors. Br J Dermatol. 2003; 149(6): 1207-1213.
- 15. Hamilton JB. Patterned loss of hair in man: Types and incidence. Ann N Y Acad Sci. 1951;53:708–728.
- 16. Montopoli M, Zumerle S, Vettor R, Rugge M, Zorzi M, Catapano CV, Carbone GM, Cavalli A, Pagano F, Ragazzi E, Prayer-Galetti T, Alimonti A, Androgen-deprivation



therapies for prostate cancer and risk of infection by SARS-CoV-2: a population-based study (n=4532), Annals of Oncology (2020), doi: <a href="https://doi.org/10.1016/j.annonc.2020.04.479">https://doi.org/10.1016/j.annonc.2020.04.479</a>
17. Goren A, Wambier CG, Herrera S, McCoy J, Vaño-Galván S, Gioia F, Comeche B, Ron R, Serrano-Villar S, Ramos PM, Cadegiani FA, Kovacevic M, Tosti A, Shapiro J, Sinclair R. Anti-androgens may protect against severe COVID-19 outcomes: results from a prospective cohort study of 77 hospitalized men. J Eur Acad Dermatol Venereol. 2020 Sep 25:10.1111/jdv.16953. doi: 10.1111/jdv.16953. Epub ahead of print. PMID: 32977363; PMCID: PMC7536996.

18. McCoy J, Cadegiani FA, Wambier CG, Herrera S, Vaño-Galván S, Mesinkovska NA, Ramos PM, Shapiro J, Sinclair R, Tosti A, Goren A. 5-Alpha-Reductase Inhibitors are Associated with Reduced Frequency of COVID-19 Symptoms in Males with Androgenetic Alopecia. J Eur Acad Dermatol Venereol. 2020 Nov 2. doi: 10.1111/jdv.17021. Epub ahead of print. PMID: 33135263.

19. Zhou T, Xu W, Zhang W, Sun Y, Yan H, Gao X, Wang F, Zhou Q, Hou J, Ren S, Yang Q, Yang B, Xu C, Zhou Q, Wang M, Chen C, Sun Y. Preclinical profile and phase I clinical trial of a novel androgen receptor antagonist GT0918 in castration-resistant prostate cancer. Eur J Cancer. 2020 Jul;134:29-40. doi: 10.1016/j.ejca.2020.04.013. Epub 2020 May 24. PMID: 32460179.

20. Wu, Siqi and Miao, Liyan and Zhou, Qianxiang and Gao, Chang and Liu, Jialin and Zhan, Qingyuan and Guo, Binbin and Li, Fang and Wang, Yirong and Xu, Hongyang and Yan, Honghua and Wu, Rui and Zhang, Shenghua and Zheng, Jiangnan and Yang, Jianfei and Wang, Shanshan and Yu, Wenkui and Niu, Haitao and Li, Fengyuan and Yang, Ling and Huang, Jianan and Lu, Xiaoting and Chen, Jiahao and Tong, Youzhi and Ma, Liandong and Zhou, Yifeng and Guo, Qiang, Suppression of Androgen Receptor (AR)-ACE2/TMPRSS2 Axis by AR Antagonists May Be Therapeutically Beneficial for Male COVID-19 Patients (April 20, 2020). Available at

SSRN: <a href="https://ssrn.com/abstract=3580526">https://ssrn.com/abstract=3580526</a> or <a href="https://dx.doi.org/10.2139/ssrn.3580526">https://dx.doi.org/10.2139/ssrn.3580526</a>

# 2. Trial Objectives

The primary purpose of this study is to evaluate the efficacy of Proxalutamide as a treatment for hospitalized COVID-19 male and female patients.

# 3. Trial Design

# 3.1 Primary Study Endpoints/Secondary Endpoints

## **Primary Outcome Measure:**

1. Treatment efficacy of Proxalutamide relative to placebo arm as assessed by the COVID-19 ordinal scale (defined in Section 5.1) [Time Frame: Day 14]

#### **Secondary Outcome Measures:**



- 1. Treatment efficacy of Proxalutamide relative to placebo arm as assessed by the COVID-19 ordinal scale (defined in Section 5.1) [Time Frame: Day 28]
- 2. Time to recovery [Time Frame: Day 1 through Day 28]
  Recovery is defined as the first day on which the subject satisfies one of the following two categories from the ordinal scale (defined in Section 5.1): 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
- 3. Proportion of death [Time Frame: Day 1 through Day 28]
  Defined as the number of subjects who have died in each arm divided by the numbers of subjects randomized to the treatment arm
- 4. Duration of new oxygen use [Time Frame: Day 1 through Day 28 ]
  Duration of new oxygen use measured in days among subjects that did not require oxygen upon randomization.
- 5. Proportion of subjects testing positive for SARS-CoV-2 [Time Frame: Day 14] Defined as the proportion of subjects in each arm with a qualitative positive rtPCR SARS-CoV-2 test from upper respiratory tract specimens

## 3.2 Study Design/Type

This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study. The study will have 2 cohorts: men and women and 2 arms:

Arm 1: Subjects administered Proxalutamide 300mg q.d for 14 days + standard of care as determined by the PI at the site

Arm 2: Subjects administered Proxalutamide placebo 300mg q.d for 14 days + standard of care as determined by the PI at the site

#### **Study Environment:**

This is a multi-center study to be conducted at multiple hospitals (the sites). This exact protocol will be followed during the study. There will be one or more PIs. The study will be approved by the appropriate Ethics Committees (IRBs). Data collection will be performed at each site by study personnel under the supervision of the PI.

#### **Study Design:**

Phase I: Enrollment (within 5 days of admission to hospital):

1. Each subject will be evaluated for the inclusion and exclusion criteria



- 2. Each subject will undergo a physical examination
- 3. Each subject (or legally authorized representative) will complete and sign the Informed Consent Form
- 4. Each subject will be assigned a subject study number
- 5. Each subject will be randomly assigned to an Arm (Section 3.3)
- 6. Based on the Arm assignment, each subject will be administered the intervention
- 7. All information will be recorded in the appropriate CRFs

#### Phase II: Outcome Assessment at Site (days 1-28):

- 1. Each subject will be evaluated daily by the PI for the outcomes of this study
- 2. Based on the Arm assignment, each subject will be administered the intervention
- 3. The PI will assess each subject for any treatment related adverse events
- 4. All information will be recorded in the appropriate CRFs

#### 3.3 Randomization

During the enrollment phase (admission to hospital), each subject will be assigned a subject study number. The first subject will be assigned the number 001 and each subject thereafter will be assigned a consecutive number i.e., 002, 003, etc.

In each cohort, subjects will be randomized into 1 of 2 arms in a 1:1 ratio each receiving an interventional treatment.

Arm 1: Subjects administered Proxalutamide 300mg q.d for 14 days + standard of care as determined by the PI at the site

Arm 2: Subjects administered Proxalutamide placebo 300mg q.d for 14 days + standard of care as determined by the PI at the site

In each cohort, each subject will be randomized using an interactive web software: Randomizer.at. The blinding table layout will be a single block. The randomization method used will be permuted blocks of size 4.

This is a blinded study. Neither participants, nor investigators, nor the study team will be aware of treatment assignments prior to the final data base locks at the conclusion of the study (or the interim analysis).




#### 3.4 Records

Each subject will be assigned a number. The numbers will be consecutive starting at 001.

A record will be created for each subject. Each record will contain a medical history, and the subject's efficacy parameters copied from the subject's charts and documented in the appropriate CRF.

The subjects' records will be stored and handled in the same manner as the PI's other clinical study patients' records are stored i.e., in a locked research storage area.

No other data will be recorded. No personal information will be kept outside the study site.

Data compiled at the end of the study will not include any information that can be used to identify individuals.

#### 3.5 Duration

The duration of the study is 28 days. There will be no study related follow-up treatment.

#### 3.6 Discontinuation

In the event that a subject experiences a SAE or an AE grade 3 or 4 (defined in Section 6) we will discontinue the study for that particular subject.

In the event a subject in any arm experiences a SAE defined as death not due to respiratory failure (presents with clear lung CT and no ARDS symptoms) the study will be discontinued. The reminder of the study shall continue.

# 3.7 Product Accountability

All interventional treatments for this study will be stored and monitored according to each hospital standard protocol.

# 3.8 Data Identification

The subject records kept by the PI will be stored and handled in the same manner as the PI's other clinical research subject records. Only authorized personnel named in this study, or medical professional retained by the PI in case of an adverse event, will have access to the subject records.

No other data will be recorded. No personal information will be kept outside the study site.

Data compiled at the end of the study will not include any information that can be used to identify individuals.



# 4. Selection and Withdrawal of Subjects

#### 4.1 Inclusion Criteria

- 1. Admitted to the hospital with symptoms of COVID-19
- 2. Male and females age ≥18 years old
- 3. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization or confirmed lung involvement by CT scan
- 4. Clinical status on the COVID-19 Ordinal Scale (defined in Section 5.1) of 3 to 6
- 5. Coagulation: INR  $\leq 1.5 \times ULN$ , and APTT  $\leq 1.5 \times ULN$
- 6. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
- 7. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

#### 4.2 Exclusion Criteria

- 1. Subject enrolled in a study to investigate a treatment for COVID-19
- 2. Requires mechanical ventilation
- 3. Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc...
- 4. Patients who are allergic to the investigational product or similar drugs (or any excipients);
- 5. Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
- 6. Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
- 7. Subjects with uncontrolled medical conditions that could compromise participation in the study(e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
- 8. Known diagnosis of human immunodeficiency virus(HIV), hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory)
- 9. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
- 10. Estimated glomerular filtration rate (eGFR) < 30 ml/min
- 11. Severe kidney disease requiring dialysis
- 12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception, as shown below, throughout the study and for 3 months after stopping GT0918 treatment. Highly effective contraception methods include:
  - Total Abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception, or



- Use of one of the following combinations (a+b or a+c or b+c):
  - a: Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
  - b: Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  - c: Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
- Female sterilization (have had prior surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment;
- Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient;
- In case of use of oral contraception women should have been stable for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment, is she considered not of child bearing potential;
- 13. Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping GT0918 treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
- 14. Subject likely to transfer to another hospital within the next 28 days
- 15. Subject (or legally authorized representative) not willing or unable to provide informed consent

# 4.3 Subject Withdrawal

Subjects may withdraw at any time for any reason. In the event the principal investigator or the site monitor believes a subject is at risk of injury the subject will be withdrawn from the study and:

- (a) If the subject has not completed the study
- (b) The subject will be replaced with another subject



- (c) The PI will follow-up with the subject every day for 14 days
- (d) The information will be reported in the appropriate CRF

## 4.4 Treatment of Subjects

Once enrolled in the study, the PI or the PI's assistant will administer the assigned treatment on a daily basis at the hospital site.

#### 4.5 Medication

Proxalutamide showed no significant inhibition on CYP1A2 and CYP2E1, weak inhibition on CYP2D6, CYP2C9, CYP2C19 and CYP3A (midazolam), but obvious inhibition on CYP3A4 (testosterone). Potential inducer on CYP3A4 at a concentration of 10μM. No inductive effects on CYP1A2 and CYP2B6 were observed in the level of enzymatic activity. Co-administration of strong/moderate CYP3A4 inducer, strong/moderate CYP3A4 inhibitor, sensitive CYP3A4/ CYP2D6 substrates and narrow therapeutic index with Proxalutamide should be used cautiously (See Appendix 1).

Note: No interaction has been reported between Proxalutamide, Nitazoxanide, and azithromycin.

Therapy prior to enrollment with any other treatment for COVID-19 or the SARS-CoV-2 infection are permitted but must be discontinued on enrollment. There is no waiting period between discontinuation of these treatments and administration of the study intervention; however, these prior treatments and their end date should be documented in the Concomitant Medication CRF.

# 4.6 Monitoring for subject compliance

The PI will monitor each subject's chart to assure daily administration of the treatment by the study staff.

# 5 Assessment of Efficacy

# 5.1 Efficacy Parameters

The following efficacy parameters will be assessed and recorded in the CRF.

#### I. COVID-19 Ordinal Scale:

The ordinal scale is an assessment of the clinical status of each subject. The scale is defined as follows:

- 8. Death:
- 7. Hospitalized, on invasive mechanical ventilation or ECMO;
- 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
- 5. Hospitalized, requiring supplemental oxygen;



- 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise;
- 3. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care;
- 2. Not hospitalized, limitation on activities;
- 1. Not hospitalized, no limitations on activities

## **II. Time to Recovery:**

Time to recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale (defined in Section 5.1): 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; or 1) Not hospitalized, no limitations on activities.

# III. "Multiple Combined Sensitive Outcome Detect Method" (combining items I and II):

- (WHO COVID ORDINAL OUTCOMES SCALE):
   a. 1 dia; b: 2 dias; c. 3 dias; d. 7 dias; e. 14 dias; f. 21 dias; g. 30 dias (cuja escala é plenamente contemplada por alguns dos desfechos descritos abaixo)
- 2. TEMPO ATÉ RECURAÇÃO regressão aos níveis 1 e 2 da WHO COVID Ordinal Outcomes Scale (dias)
- 3. POSITIVIDADE DA rtPCR-SARS-CoV-2 a. 7 dias; b. 14 dias; c. 30 dias (%)
- 4. TEMPO ATÉ REMISSÃO DE CADA SINTOMA (dias)
- 5. TEMPO ATÉ REMISSÃO COMPLETA DOS SINTOMAS (dias)
- 6. TEMPO ATÉ RECUPERAÇÃO DA CAPACIDADE DE REALIZAÇÃO DE ATIVIDADES DIÁRIAS DEVIDO AOS SINTOMAS DE COVID-19 (Nível 1 da WHO COVID Ordinal Outcomes Scale) (dias)
- 7. NECESSIDADE DE UNIDADE INTENSIVA (%)
- 8. NECESSIDADE DE VENTILAÇÃO MECÂNICA (%)
- 9. TEMPO DE HOSPITALIZAÇÃO (dias)
- 10. TEMPO DE OXIGENIOTERAPIA (dias) (se necessário)
- 11. TEMPO DE UNIDADE DE TERAPIA INTENSIVA (dias) (se necessário)
- 12. TEMPO DE VENTILAÇÃO MECÂNICA (dias) (se necessário)
- 13. NECESSIDADE DE USO DE VASOATIVOS (%)
- 14. MORTE (%)

# 5.2 Method and Timing

For each study day while the subject is hospitalized, the PI will record the clinical assessment on an 8- point ordinal scale as follows:

• Day 1 – The clinical assessment at the time of enrollment.




- Day 2 The most severe clinical assessment occurring any time between enrollment and midnight the day following enrollment.
- Day 3-28 (or until discharged) The most severe assessment occurring from midnight to midnight of the prior day (e.g., the value recorded on Day 3 will be the most severe outcome that occurred on Day 2).

If the subject is no longer hospitalized at day 28, a clinical assessment will be made by an inperson or phone visit; otherwise, it would be recorded as missing data.

## 6 Assessment of Safety

## 6.1 Safety Parameters

Safety parameters will be assessed as follows:

## **I. Physical Examination:**

The PI will conduct a thorough physical examination during screening. The assessment will be recorded in the appropriate CRF.

## **II. Clinical Laboratory Evaluations:**

The following tests will be conducted: WBC, differential, Hgb, PLT, creatinine, glucose, total bilirubin, AST, ALT and coagulation PT.

### **III. Adverse Events:**

Safety will be assessed by summarizing the incidence and type of Adverse Events in a CRF form.

## 6.2 Method and Timing

The assessments, as described in section 6.1, will occur as follows:

## **I. Physical Examination**

The assessment will occur at screening. The information will be recorded in the appropriate CRF.

### **II. Clinical Laboratory Evaluations:**

The assessment will occur upon admission to the hospital as well as at day 14. Additional laboratory tests or timing may be ordered as deemed necessary by the PI.

#### **III. Adverse Events:**

Adverse events will be assessed daily during the 28 day duration of the trial. The information will be recorded in the appropriate CRF.

The methods employed for completing assessments are described in section 6.1


This material is the property of the Applied Biology Inc. Do not disclose or use except as authorized.



## 6.3 Adverse Events

## **6.3.1** Definition of Adverse Event (AE)

AE means any medical event associated with the use of an intervention, whether or not considered intervention-related. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product.

Any medical condition that is present at the time that the subject is screened will be considered as baseline and not reported as an AE. However, if the severity of any pre-existing medical condition increases, it should be recorded as an AE.

Given the nature of severity of the underlying illness, subjects will have many symptoms and abnormalities in vitals and laboratory. All Grade 3 and 4 AEs will be captured as AEs in this trial.

## 6.3.2 Definition of Serious Adverse Event (SAE)

An SAE is defined as "An AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in any of the following outcomes: Death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse." "Lifethreatening" refers to an AE that at occurrence represents an immediate risk of death to a subject. An event that may cause death if it occurs in a more severe form is not considered life-threatening. Similarly, a hospital admission for an elective procedure is not considered a SAE. All SAEs, as with any AE, will be assessed for severity and relationship to study intervention. All SAEs will be recorded on the appropriate SAE CRF. All SAEs will be followed through resolution or stabilization by a licensed study physician (for IND studies, a physician listed on the Form FDA 1572 as the site PI or Sub-Investigator). All SAEs will be reviewed and evaluated by DMID and will be sent to the SMC (for periodic review), and the IRB/IEC.

### 6.3.3 Suspected Unexpected Serious Adverse Reactions (SUSAR)



A SUSAR is any SAE where a causal relationship with the study product is at least reasonably possible but is not listed in the Investigator Brochure (IB), Package Insert, and/or Summary of Product Characteristics.

### 6.3.4 Classification of an Adverse Event

The determination of seriousness, severity, and causality will be made by an on-site investigator who is qualified (licensed) to diagnose AE information, provide a medical evaluation of AEs, and classify AEs based upon medical judgment. This includes but is not limited to physicians, physician assistants, and nurse practitioners.

## **6.3.5** Severity of Adverse Events

All AEs and SAEs will be assessed for severity, according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 2.1 (July 2017). For AEs not included in the protocol defined grading system, the following guidelines will be used to describe severity.

Mild (Grade 1): Events that are usually transient and may require only minimal or no treatment or therapeutic intervention and generally do not interfere with the subject's usual activities of daily living.

Moderate (Grade 2): Events that are usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research subject.

Severe (Grade 3): Events interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating.

Severe (Grade 4): Events that are potentially life threatening.

AEs characterized as intermittent require documentation of onset and duration of each episode. The start and stop Duration of each reported AE will be recorded on the appropriate CRF. Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of intensity.

### **6.3.6** Relationship to Study Intervention

For each reported adverse reaction, the PI or designee must assess the relationship of the event to the study product using the following guideline:

Related – The AE is known to occur with the study intervention, there is a reasonable possibility that the study intervention caused the AE, or there is a temporal relationship between the study intervention and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study intervention and the AE.



Not Related – There is not a reasonable possibility that the administration of the study intervention caused the event, there is no temporal relationship between the study intervention and event onset, or an alternate etiology has been established.

## 6.3.7 Time Period and Frequency for Event Assessment and Follow-Up

For this study, all Grade 3 and 4 AEs and all SAEs occurring from the time the informed consent is signed through the Day 28 (end of study) visit will be documented, recorded, and reported.

## 6.3.8 Investigators Reporting of AEs

Information on all AEs should be recorded on the appropriate CRF. All clearly related signs, symptoms, and results of diagnostic procedures performed because of an AE should be grouped together and recorded as a single diagnosis. If the AE is a laboratory abnormality that is part of a clinical condition or syndrome, it should be recorded as the syndrome or diagnosis rather than the individual laboratory abnormality. Each AE will also be described in terms of duration (start and stop date), severity, association with the study product, action(s) taken, and outcome.

## 6.3.9 Serious Adverse Event Reporting

### 6.3.9.1 Investigators Reporting of SAEs

Any AE that meets a protocol-defined criterion as a SAE must be submitted immediately (within 24 hours of site awareness) on an SAE form to the DMID Pharmacovigilance Group, at the following address:

DMID Pharmacovigilance Group

Clinical Research Operations and Management Support (CROMS)

6500 Rock Spring Dr. Suite 650

Bethesda, MD 20817, USA

SAE Hot Line: 1-800-537-9979 (US) or 1-301-897-1709 (outside US) SAE FAX Number: 1-800-275-7619 (US) or 1-301-897-1710 (outside US) SAE Email Address:

PVG@dmidcroms.com

Other supporting documentation of the event may be requested by the DMID Pharmacovigilance Group and should be provided as soon as possible. The DMID Medical Monitor will review and assess the SAE for regulatory reporting and potential impact on study subject safety and protocol conduct. At any time after completion of the study, if the site PI or appropriate sub-investigator becomes aware of an SAE, the site PI or appropriate sub-investigator will report the event to the DMID Pharmacovigilance Group.

### 6.3.9.2 Regulatory Reporting of SAEs



Following notification from the site PI or appropriate sub-investigator, DMID, as the IND sponsor, will report any SUSAR in an IND safety report to the FDA and will notify all participating site PIs as soon as possible. DMID will report to the FDA any unexpected fatal or life-threatening suspected adverse reaction as soon as possible, but in no case later than 7 calendar days after the sponsor's initial receipt of the information. If the event is not fatal or life- threatening, the IND safety report will be submitted within 15 calendar days after the sponsor determines that the information qualifies for reporting as specified in 21 CFR Part 312.32. Relevant follow up information to an IND safety report will be submitted as soon as the information is available. Upon request from FDA, DMID will submit to the FDA any additional data or information that the agency deems necessary, as soon as possible, but in no case later than 15 calendar days after receiving the request. SAEs that are not SUSARs will be reported to the FDA at least annually in a summary format which includes all SAEs. Sites may have additional local reporting requirements (to the IRB and/or national regulatory authority).

## **6.3.10** Reporting Events to Subjects

Subjects will be informed of any severe AEs or SAEs that occur as part of their participation in this trial.

## **6.3.11** Reporting of Pregnancy

Pregnancy is not defined as an AE. However, any pregnancy that occurs during study participation should be reported to the sponsor on the appropriate CRF. Pregnancy should be followed to outcome.

## 6.4 Unanticipated Problems

### 6.4.1 Definition of Unanticipated Problems (UP)

An Unanticipated Problem is any event, incident, experience, or outcome that meets the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied;
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

### 6.4.2 Unanticipated Problem Reporting



To satisfy the requirement for prompt reporting, unanticipated problems (UP) will be reported using the following timeline: UPs that are SAEs will be reported to the IRB and to the Statistical and Data Coordinating Center (SDCC)/study sponsor within 24 hours of the investigator becoming aware of the event per the above describe SAE reporting process. Any other UP will be reported to the IRB and to the SDCC/study sponsor within 3 days of the investigator becoming aware of the problem.

## 6.4.3 Reporting Unanticipated Problems to Subjects

Subjects will be informed of any UPs that occur as part of their participation in this trial.

## 7 Statistical Plan

## 7.1 Statistical Methods

## I. General Principles:

- Double-blinded, placebo controlled randomized interventional study with a two-sided type I error rate of 0.05.
- Continuous variables will be expressed as median (interquartile range [IQR]) and categorical variables will be expressed as a number
- 95% confidence intervals will be calculated for the primary outcome
- Group comparisons will be analyzed by the Wilcoxon rank sum test or  $\chi 2$  test
- The placebo arm will be used as a reference group when calculating treatment effects
- Differences between rates of clinical improvement will be calculated using unadjusted ordinal logistic regression or Cox proportional hazard models
- Statistical analyses will be conducted using XLSTAT version 2020.5.1 (Addinsoft, Inc.)

### **II. Statistical Hypotheses:**

The primary endpoint is the distribution of clinical assessments on the COVD-19 ordinal scale at day 14. The primary outcome will be analyzed using the Wilcoxon rank sum test.

The Null Hypothesis (H<sub>0</sub>) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with Proxalutamide is equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with the Proxalutamide placebo

The Alternative Hypothesis (H<sub>A</sub>) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with Proxalutamide is not equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with the Proxalutamide placebo



Mathematically written as:

$$H_0: P(X > Y) = P(Y > X)$$

$$H_A: P(X > Y) \neq P(Y > X)$$

Where X and Y are randomly selected clinical assessments from the two treatment arms in the study.

## **III. Primary Efficacy Analysis:**

- The non-parametric Wilcoxon rank sum test (Mann Whitney U) will be used to assess the primary end point.
- P-values <0.05 will be considered significant. All statistical analysis will be based on the intent-to-treat (ITT) population. All missing data will be described.

## 7.2 Sample Size Estimates

## **Assumptions:**

- The sample size estimation is based on the results reported in the placebo arm of the Adaptive COVID-19 Treatment Trial (NCT04280705)
- On day 15, 61% of subjects in NCT04280705 placebo group remained hospitalized.
- The odds ratio of improvement in the ordinal scale in the Proxalutamide arm compared to the Proxalutamide placebo is at least 2.0
- The study has two arms with randomization at 1:1 ratio
- 90% power to detect an odds ratio of 2.0 using a two-tailed test with a type I error rate of 5%
- According to NCT04280705 protocol "The sample size to detect a given odds ratio for 1:1 randomization using a 2-tailed test at level  $\alpha$  is estimated by the equation below.  $\lambda$  is the log odds ratio, pi is the overall probability (combined over both arms) of being in the ith category of the K ordinal outcomes, and  $z\alpha/2$  and  $z\beta$  are the  $1 \alpha/2$  and  $1 \beta$  quantiles of the standard normal distribution."

$$\frac{12(z_{\alpha/2} + z_{\beta})^{2}}{\lambda^{2}(1 - \sum_{i=1}^{K} p_{i}^{3})'}$$

- The estimated distribution is based on NCT04280705 protocol scenario 4
- 3.5% of the subjects will not complete the study based on NCT04280705

## Sample Size Estimate:



Based on the assumptions above, we calculated that at a minimum we would need to recruit for each cohort 294 subjects (147 subjects in each arm) i.e., a total of approximately 600 subjects.

## 7.3 Subject Population(s) for Analysis

- The primary analysis will be based on the intent-to-treat (ITT) population. The data from all subjects enrolled in the study will be analyzed.
- The safety analysis will be based on a modified intent-to-treat (MITT) population i.e., subjects who received at least one dosage of the interventional treatment.
- Subgroup analysis based on: 1) age stratification; and 2) androgen status as defined by the "Gabrin sign" or "PCOS signs" will be conducted for the primary and secondary outcomes.

## 7.4 Interim Analysis

Interim efficacy and safety data will be made upon recruitment of 50% of the subjects.

## 7.5 Termination Criteria

Upon occurrence of any one of the events listed below, the study will terminate or be modified accordingly:

- Completion of the study by a sufficient number of subjects (294 subjects) to reach our confidence level
- Termination of Arm 1: Serious adverse event due to treatment with Proxalutamide
- Substantial evidence of treatment difference between the arms. The study design will be modified to an open-label study.

## 7.6 Accountability Procedure

The data will be analyzed by a bio-statistics expert. The data will also be independently verified by an outside expert consultant.

## 7.7 Deviation Reporting

No deviation from the plan will be implemented without the prior review and approval of the EC/IRB.

## 8 Direct Access to Source Data/Documentation

The PI and hospital will permit trial-related monitoring, audits, IRB/IEC(s) review and regulatory inspection(s) by providing direct access to source data/documentation.



## 9 Quality Control and Quality Assurance

Every effort will be made to keep staff assignments consistent throughout the entire study. The PI who assesses the subject at baseline should follow the subject throughout the completion of the study. This will ensure that this study is conducted – and that data is generated, documented (recorded), and reported - in compliance with this protocol, with GCP, and any other applicable regulatory requirements. The study monitor will audit the study procedures and CRFs throughout the study.

## 10 Ethical Considerations

This study will be conducted according to US and international standards of Good Clinical Practice (FDA regulations 21 CFR 312 for IND studies and FDA guidance E6) for all studies. Applicable government regulations and hospital research policies and procedures will also be followed.

This protocol and any amendments will be submitted to the Institutional Review Board (IRB) for formal approval to conduct the study. The decision of the IRB concerning the conduct of the study will be made in writing to the investigator.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB. The formal consent of a subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. This consent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

## 11 Data Handling and Record Keeping

During enrollment, each subject will be assigned a number. The numbers will be consecutive starting at 001.

During enrollment a record will be created for each subject. Each record will contain the subject's demographics, subject's efficacy parameters and any adverse events or study related information.

The subjects' records will be stored and handled in the same manner as the PI's patients' records.

The study monitor will keep a separate record at the monitor's office of each subject's identification number, the treatment administered to the subject (arm assignment), outcomes and any laboratory results.

No other data will be recorded. No personal information will be kept outside the study site.



Data compiled at the end of the study will not include any information that can be used to identify individuals.

The site will keep all subject records for a minimum of 3 years after the completion of the study.

## 12 Finance and Insurance

The Principal Investigator will be responsible for the cost of study. The site carries insurance for accidental injury. There is no other insurance.



## APPENDIX 1

## Drugs that should be used cautiously with Proxalutamide

## Strong CYP3A4 inducer

Avamibe, Carbamazepine, Phenytoin, Rifampicin, Mitotan, Nevirapine, Phenobarbital, Rifabutin, Rifapentine, St. John's wort, Alfentanil, Ryclosporin, Dihydroergotamine / Ergotamine, Fentanyl, Irinotecan, Pimozit, Quinidine, Sirolimus, Tacrolimus

## Moderate CYP3A4 inducer

Smacet, Tavern, Bosentan, Efaviron, Etruverin, Lopinavir, Modafinil, Nafcillin, Thalidazine, Tiranavir, Ritonavir

## Strong CYP3A4 inhibitor

Posidovir, Clarithromycin, Conivatan, Indinavir, Itraconazole, Ketoconazole, lopinavir / Ritonavir, Mibedil, Nefazodone, Nefenavir, Posaconazole, Ritonavir, Saquinavir, Trapivir, Taliomycin, Voriconazole, Etigavir / Ritonavir, Fluconazole, Tiranavir / Ritonavir, Acetamycin

### **Moderate CYP3A4 inhibitors**

Apronavir, Aripitan, Azanavir, Casopitam, Cimetidine, Ciprofloxacin, Clazotinib, Cyclosporin, Dalunavir, Diltiazem, Dronedarone, Erythromycin, Imatinib, Tofesoyang, Verapamil

### Sensitive CYP3A4 substrates

Remifentanil, Aripiptam, Budesonide, Buspirone, Conivatan, Daphnesin, Darunavir, Dasatinib, Dronedarone, Eletroptan, Eplerenone, Everolimus, Felodipine, Indinavir, Fluticasone, Lopinavir, Lovastatin, Lulasidone, Maravelo, Midazolam, Nisoldipine, Quetiapine, Saquinavir, Sildenafil, Simvastatin, Sirolimus, Tolvaptan, Tiranavir, Triazolam, Vardenafil

## Narrow therapeutic index CYP3A4 Substrate

Astemizole, Cisapride, Cyclosporine, Dihydroergotamine, Fentanyl, Pethidine, Quinidine, Tacrolimus, Terfenadine

#### Sensitive CYP2D6 substrates

Tomoxetine, Decipamine, Dextromethorphan, Metoprolol, Nebeprolol, Perphenazine, Tolterodine, Venlafaxine, Avamibe, Carbamazepine, Phenytoin sodium, Rifampicin




# Narrow therapeutic index CYP2D6 Substrate

Thioridazine



| Revision History | | | | |
|---|---|---|---|---|
| Revision | Description of Change | | Date | Signature |
| 1 | New draft release | Andy Goren | Dec 27, 2020 | |
| 2 | Amendments to end points | Andy Goren | Dec 29, 2020 | |
| 3 | Amended AE section | Andy Goren | Dec 30, 2020 | |
| 4 | Amended to include female cohort | Flavio Cadegiani | Jan 10, 2021 | |
| 5 | Final review for female cohort | Andy Goren | Jan 10. 2021 | |
| 6 | Added exclusions for sexual activity and minor corrections | Andy Goren | Jan 11, 2021 | = |
| 7 | Changed randomization model | Andy Goren | Jan 19, 2021 | |
| 8 | Amended inclusion criteria | Andy Goren | February 1, 2021 | |

# FINAL STATISTICAL PLAN WITH SUMMARY OF CHANGES FROM THE FINAL PROTOCOL

We had to make minor adjustments to the statistical plan of the final protocol while writing the manuscript to make the statistical plan more stringent and clearer. The rationale for each change or no change is also presented.

## **Table of contents:**

| 1. | Primary Outcome Measure | . 1 |
|----|----------------------------|-----|
| 2. | Secondary Outcome Measures | . 2 |
| 3. | General principles | . 4 |
| 4. | Statistical hypothesis | . 5 |
| 5. | Primary analysis efficacy | . 6 |
| 6. | Sample size calculation | . 7 |

# 1. Primary Outcome Measure

| Proposed in the final protocol | Final statistical Plan | Rationale |
|---|---|---|
| Treatment efficacy of | No change | The distribution analysis of all the |
| proxalutamide relative to | | COVID-19 8-point ordinal scale scores |
| placebo arm as assessed by the | | at day 14 covers all possible scores, 1 |
| COVID-19 ordinal scale [time | | to 8. This is better illustrated |
| frame: day 14] | | graphically for group comparison. |
| No specific measure of effect | Recovery ratio was defined as | Scores 1-2 represent a clear cut for |
| was appointed for the Primary | the measure of effect for the | recovery (alive hospital discharge). |
| efficacy analysis (quantitative | primary outcome. The treatment | |
| efficacy measure). | efficacy of proxalutamide was | |
| | assessed by the proportion of | |
| | recovered patients in both study | |
| | arms [time frame: 14 days]. | |
| | Recovery was defined as | |
| | reaching scores 1 and 2 in the | |
| | COVID-19 ordinal scale | |

# 2. Secondary Outcome Measures

| As proposed in the final protocol | Done in the final statistical Plan | Rationale |
|---|---|---|
| Treatment efficacy of Proxalutamide relative to placebo arm as assessed by the COVID- 19 ordinal scale (defined in Section 5.1) [Time Frame: Day 28] | A clear cut-off point was used in the COVID-19 scale (scores 1 and 2) so that we were able to measure the effect size <b>recovery ratio</b> [time frame: 28 days]. | All scores at Day 28 are informative and is better presented in a graph. As reported for the primary outcome, we clarified a measure of effect within this secondary outcome measure. |
| Time to recovery [Time Frame: Day 1 through Day 28] Recovery is defined as the first day on which the subject satisfies one of the following two categories from the ordinal scale.1): 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. | Name changed to post-randomization time to recover/alive hospital discharge [time frame: day 1 to day 28] in median days (interquartile range). Recovery was defined as the first day on which the subject reached scores 1 and 2 in the COVID-19 ordinal scale. | We needed to be more specific in this outcome to make it clearer and reproducible. |
| Proportion of death [Time Frame: Day 1 through Day 28] Defined as the number of subjects who have died in each arm divided by the numbers of subjects randomized to the treatment arm | Name changed to 28-day all-cause mortality rate. The proportion of patients who reached score 8 in the 19-COVID ordinal scale after randomization. [Time frame: 28 days] | The outcome is still the same described in the statistical plan of the final protocol, however we just clarified that it refers to all-cause mortality. All-cause mortality is a more stringent measure, and therefore this change goes against the direction of the bias. Although mortality at 14 days could be contemplated in the original Primary outcome (score 8), we decided to analyze mortality at 28 days only, which is more stringent and reflects the intention-to-treat. |
| Duration of new oxygen use<br>[Time Frame: Day 1 through<br>Day 28] | Excluded | This outcome measure was not adequately reported by the hospital sites, and therefore we have not included it in the final statistical plan. |
| Proportion of subjects testing positive for SARS-CoV-2 [Time Frame: Day 14] | Excluded | This outcome also needed to be abandoned because we lacked financial resources to test all patients again for SARS-CoV-2 at day 14. |
| Subgroup analysis based on: 1) age stratification; and 2) androgen status as defined by "Gabrin sign" or "PCOS signs" will be conducted for the primary and secondary outcomes. | Changed to include the subgroup analysis per 1) baseline score (severity of the disease), 2) gender and 3) hospital site. No hypothesis testing was performed in these subgroup analyses to avoid finding significant p-values by chance due to multiple comparisons. Androgen status was excluded from the subgroup analysis. | Several reasons led us to make these new subgroup analyses: 1. Age was lower than expected, lower age cut-offs did not show relevant findings to be reported, possibly in the future we may plan for a multivariate analysis with factors such as women post-menopause. Also, pre-determining age cut-offs for analyses were needed. Age |

- distribution graphs were included in the supplement.
- 2. Since the randomization scheme was changed in the small hospital located in the remote Amazon areas to control for sharing and unblinding in these regions (see randomization details in the supplement), we needed to evaluate if there was interaction between the overall effect size [recovery ratio, and all-cause mortality ratio] per city of sites. Important to say here that in the hospital centers located in the capital of the state of Amazonas, randomization scheme was performed as planned.
- 3. Since men are by definition more androgenic it was important to evaluate the effects specifically.
- 4. Finally, we checked if there were an interaction effect between the patients with more severe presentations such as baseline score 6 compared to 5, 4,

# 3. General principles

| As proposed in the final protocol | Done in the final statistical Plan | Rationale |
|---|---|---|
| Continuous variables will be expressed as median (interquartile range [IQR]) and categorical variables will be expressed as a number | Continuous variables were expressed as median (IQR) and categorical variables were expressed as a number and in a risk percentage. | Expression of the categorical variables only as a number is not sufficient to allow for calculation of risk ratios. Then, absolute risk ratios were calculated for primary (14-day Overall Recovery rate) and secondary outcomes (28-day recovery rate and 28-day all-cause mortality) |
| 95% confidence intervals will be calculated for the primary outcome | 95% confidence intervals will<br>be calculated for the primary<br>outcome, secondary outcomes<br>and subgroup analysis. | All secondary outcomes expressed in ratios were reported along with the 95% confidence interval to allow for a better understanding of the effect sizes. |
| Group comparisons will be analyzed by the Wilcoxon rank sum test or χ2 test | For all categorial effect sizes, hypothesis testing was performed with the χ2 test, including risk ratios. 95% Confidence intervals were reported in results tables, for the primary endpoint <b>Overall Recovery Ratio</b> ), along with the P value. For the Adverse AE table, P-values were included. Other outcomes described as median and IQR were compared with the Wilcoxon rank sum test. | The primary hypothesis testing previously stated was maintained. However, we explained in which cases the different tests were applied to increase transparency. |
| Differences between rates of clinical improvement will be calculated using unadjusted ordinal logistic regression or Cox proportional hazard models | We used Kaplan-Meier's survivor function for estimates of proportion surviving, and failure function for estimates of alive hospital discharges. Cox proportional hazards model was kept only to calculate hazard ratio (HR) for death and its 95% confidence interval (CI). Graphical assessment and Kaplan-Meier versus predicted survival showed that of the proportional-hazards assumption has not been violated | For better demonstration of the 95% CI and timeline of the evolution of the outcomes in figures. For measure of effect, as stated in the Primary and Secondary outcomes, we adopted relative risk (or Risk Ratio) for easier understanding. |
| Statistical analyses will be conducted using XLSTAT version 2020.5.1 (Addinsoft, Inc.) | Statistical analysis was conducted using Stata/SE version 16.1 for Mac (StataCorp LLC, College Station, TX, USA). | Preference of the team performing statistical analysis |

# 4. Statistical hypothesis

| As proposed in the final | Done in the final statistical | Rationale |
|---|---|---|
| | Plan | |
| protocol The primary endpoint is the distribution of clinical assessments on the COVID-19 ordinal scale at day 14. The primary outcome will be analyzed using the Wilcoxon rank sum test. | Plan The primary efficacy endpoint was described as the overall 14-day recovery ratio. This effect measure was obtained after dichotomization of the COVID-19 ordinal scale for scores 2 and 1, representing patients that were discharged from hospital. | Although the distribution is still presented graphically, and tested for statistical significance, a clear cut-off point in the COVID-19 ordinal scale was used to obtain the <b>Overall Recovery Ratio</b> . Recovery ratio is a clinically meaningful effect measure. |
| The Null Hypothesis (H0) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with Proxalutamide is equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with the Proxalutamide placebo | The null hypothesis applied to the primary endpoint <b>Overall Recovery Ratio</b> is that there is no association between the recovery risk rates of the study arms and the type of treatment (proxalutamide or placebo) in the hospitalized patients with COVID-19 | Since the primary outcome was refined with a clear efficacy endpoint, defined as a binary measure, the null hypothesis was rephrased to be in line with the chi-square test. |
| The Alternative Hypothesis (HA) is that the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with Proxalutamide is not equal to the distribution of clinical assessments on the COVD-19 ordinal scale at day 14 among hospitalized COVID-19 subjects treated with the Proxalutamide placebo | The alternative hypothesis applied to the primary endpoint <b>Overall Recovery Ratio</b> is that the there is an association between the recovery risk rates of the study arms and the type of treatment (proxalutamide or placebo) in the hospitalized patients with COVID-19, meaning that the experimental treatment may affect the <b>Overall Recovery Ratio</b> . | The primary outcome was refined with a clear efficacy endpoint, defined as a binary measure the alternative hypothesis was rephrased to be in line with the chi-square test. |

# 5. Primary analysis efficacy

| As proposed in the final | Done in the final statistical | Rationale |
|---|---|---|
| protocol | Plan | |
| The non-parametric Wilcoxon rank sum test (Mann Whitney U) will be used to assess the primary end point. P-values <0.05 will be considered significant. All statistical analysis will be based on the intent-to-treat (ITT) population. All missing data will be described. | The non-parametric Wilcoxon rank sum test was used to assess some of the secondary outcomes described above. The intention-to-treat protocol was performed in the final analysis. Missing data was reported. | The primary outcome was refined with a clear efficacy endpoint, defined as a binary measure, and thus, Wilcoxon Rank Sum test was not appropriate for such type of variable. |
| No measure of effect | Included measure of effect: Overall Recovery Ratio [time frame: 14 days] | Although we meant to calculate the overall recovery ratio, the outcome was not clearly described in the statistical plan of the protocol, and sample size was based on odds ratio for recovery. |

# 6. Sample size calculation

| As proposed in the final | Done in the final statistical<br>Plan | Rationale |
|---|---|---|
| The sample size estimation is based on the results reported in the placebo arm of the Adaptive COVID-19 Treatment Trial (NCT04280705) protocol scenario 4: On day 15, 61% of subjects in NCT04280705 placebo group remained hospitalized. For 90% power to detect an odds ratio of 2.0 using a two-tailed test with a type I error rate of 5%, and 3.5% of the subjects will not complete the study based on NCT04280705 | No change. However, we noticed that the way the sample size estimation was described may be hard for many readers to follow it. An odds ratio for improvement of 2 over a baseline recovery risk of 39% (NCT04280705, scenario 4), results in a difference of 14% in the absolute recovery rate. The sample size was calculated to be able to detect a difference of 14% in Overall Recovery Rate at 14 days (risk ratio of 1.36) with a power of 90% and a type I error of 5%, over the estimated 39% recovery rate for the placebo group, and 3.5% non-compliance/cross over in the study groups. | Although no change was done in the sample size estimate, we rewrote it using simpler and more direct terms. |
| Sample size estimate: Based on the assumptions above, we calculated that at a minimum we would need to recruit for each cohort 294 subjects (147 subjects in each arm) i.e., a total of approximately 600 subjects. | No change | We verified that the sample size was still 90% powered after inclusion of baseline score 6 to the final protocol. |

These minor changes in the statistical analysis plan were performed while writing the manuscript.

Researchers involved in the statistical analysis that implemented the changes:

Dr. Carlos Wambier, MD, PhD

Dr Alessandra Reis, DDS, PhD